CLINICAL TRIAL: NCT01991795
Title: A Multinational, Randomised, Double-Blind, Placebo-Controlled Trial to Evaluate the Effect of Ticagrelor Twice Daily on the Incidence of Cardiovascular Death, Myocardial Infarction or Stroke in Patients With Type 2 Diabetes Mellitus (THEMIS - Effect of Ticagrelor on Health Outcomes in Diabetes Mellitus Patients Intervention Study).
Brief Title: A Study Comparing Cardiovascular Effects of Ticagrelor Versus Placebo in Patients With Type 2 Diabetes Mellitus
Acronym: THEMIS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: D513BC00001
Record Dates: First submitted 2013-11-18; First posted 2013-11-25 (Estimated); Results first posted 2020-03-18 (Actual); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diabetes; Coronary artery disease; Outcome; Prevention; Antiplatelet
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Coronary Artery Disease | interventions — Ticagrelor

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ticagrelor 60 mg (Experimental): Initially ticagrelor 90 mg or corresponding placebo was the selected dose, but reduced to ticagrelor 60 mg or corresponding placebo in Clinical Study Protocol Amendment No 1.
  Interventions: Drug: Ticagrelor 60 mg
- Ticagrelor placebo (Placebo Comparator): Initially ticagrelor 90 mg or corresponding placebo was the selected dose, but reduced to ticagrelor 60 mg or corresponding placebo in Clinical Study Protocol Amendment No 1.
  Interventions: Drug: Ticagrelor placebo

INTERVENTIONS:
Drug: Ticagrelor 60 mg — Ticagrelor 60 mg bd taken orally as tablets
  Other Names: Brilinta/Brilique
  Arms: Ticagrelor 60 mg
Drug: Ticagrelor placebo — Ticagrelor placebo bd taken orally as tablets
  Arms: Ticagrelor placebo

SUMMARY:
The purpose of this study is to compare the effect of ticagrelor versus placebo in patients with Type 2 Diabetes Mellitus.

DETAILED DESCRIPTION:
A multinational, randomised, double-blind, placebo-controlled phase IIIb trial to evaluate the effect of ticagrelor twice daily on the incidence of cardiovascular death, myocardial infarction or stroke in patients with type 2 diabetes mellitus

ELIGIBILITY:
Inclusion Criteria:

Men or women ≥50 years of age with type 2 diabetes mellitus on treatment with a glucose lowering medication since at least 6 months, and either documented coronary artery occlusive disease or previous revascularization of a coronary artery.

Key Exclusion Criteria:

History of myocardial infarction or any stroke; planned treatment with agents inhibiting blood clotting; planned use of ASA/Aspirin at doses above 150 mg daily; planned coronary, cerebrovascular, or peripheral arterial revascularization; patients with known bleeding disorders and patients who need chronic oral anticoagulant therapy or chronic low-molecular-weight heparin; history of intracranial bleeding at any time, or a history of bleeding from the gastrointestinal tract within the last 6 months or a major surgery within the last 30 days; patients with known severe liver disease or with kidney failure requiring dialysis

Ages: 50 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19271 (Actual)
Dates: Start 2014-02-10 (Actual); Primary Completion 2019-01-25 (Actual); Study Completion 2019-01-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Gabriel Steg, MD, Principal Investigator — Hôpital Bichat-Claude Bernard 46 Rue Henri Huchard, Paris; Deepak L. Bhatt, MD, Principal Investigator — Brigham and Women's Hospital75 Francis Street, Boston
Locations (887):
- United States (241):
  - Research Site, Alexander City, Alabama
  - Research Site, Birmingham, Alabama
  - Research Site, Fairhope, Alabama
  - Research Site, Huntsville, Alabama
  - Research Site, Mobile, Alabama
  - Research Site, Montgomery, Alabama
  - Research Site, Sheffield, Alabama
  - Research Site, Tuscumbia, Alabama
  - Research Site, Cottonwood, Arizona
  - Research Site, Glendale, Arizona
  - Research Site, Tucson, Arizona
  - Research Site, Little Rock, Arkansas
  - Research Site, Anaheim, California
  - Research Site, Bakersfield, California
  - Research Site, Beverly Hills, California
  - Research Site, Fremont, California
  - Research Site, Fresno, California
  - Research Site, Irvine, California
  - Research Site, La Mesa, California
  - Research Site, Long Beach, California
  - Research Site, Los Alamitos, California
  - Research Site, Los Angeles, California
  - Research Site, Mission Hills, California
  - Research Site, Newport Beach, California
  - Research Site, Sacramento, California
  - Research Site, San Diego, California
  - Research Site, Stanford, California
  - Research Site, Stockton, California
  - Research Site, Tarzana, California
  - Research Site, Torrance, California
  - Research Site, Denver, Colorado
  - Research Site, Bridgeport, Connecticut
  - Research Site, Greenwich, Connecticut
  - Research Site, Bradenton, Florida
  - Research Site, Clearwater, Florida
  - Research Site, Cooper City, Florida
  - Research Site, Coral Springs, Florida
  - Research Site, Crystal River, Florida
  - Research Site, Cutler Bay, Florida
  - Research Site, Daytona Beach, Florida
  - Research Site, DeLand, Florida
  - Research Site, Fort Lauderdale, Florida
  - Research Site, Hialeah, Florida
  - Research Site, Hollywood, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, Lake Worth, Florida
  - Research Site, Largo, Florida
  - Research Site, Merritt Island, Florida
  - Research Site, Miami, Florida
  - Research Site, Miami Gardens, Florida
  - Research Site, Miami Shores, Florida
  - Research Site, Miami Springs, Florida
  - Research Site, Naples, Florida
  - Research Site, New Smyrna Beach, Florida
  - Research Site, North Miami Beach, Florida
  - Research Site, Ocala, Florida
  - Research Site, Ormond Beach, Florida
  - Research Site, Panama City, Florida
  - Research Site, Port Charlotte, Florida
  - Research Site, Saint Cloud, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Columbus, Georgia
  - Research Site, Cumming, Georgia
  - Research Site, Decatur, Georgia
  - Research Site, Gainesville, Georgia
  - Research Site, Tucker, Georgia
  - Research Site, Nampa, Idaho
  - Research Site, Arlington Heights, Illinois
  - Research Site, Chicago, Illinois
  - Research Site, Crystal Lake, Illinois
  - Research Site, Elmhurst, Illinois
  - Research Site, Evanston, Illinois
  - Research Site, Gurnee, Illinois
  - Research Site, Hinsdale, Illinois
  - Research Site, Moline, Illinois
  - Research Site, North Chicago, Illinois
  - Research Site, Peoria, Illinois
  - Research Site, Anderson, Indiana
  - Research Site, Elkhart, Indiana
  - Research Site, Fort Wayne, Indiana
  - Research Site, Greenfield, Indiana
  - Research Site, Indianapolis, Indiana
  - Research Site, Muncie, Indiana
  - Research Site, Munster, Indiana
  - Research Site, Davenport, Iowa
  - Research Site, West Des Moines, Iowa
  - Research Site, Wichita, Kansas
  - Research Site, Crestview Hills, Kentucky
  - Research Site, Owensboro, Kentucky
  - Research Site, Alexandria, Louisiana
  - Research Site, Bossier City, Louisiana
  - Research Site, Covington, Louisiana
  - Research Site, Crowley, Louisiana
  - Research Site, Minden, Louisiana
  - Research Site, Monroe, Louisiana
  - Research Site, Shreveport, Louisiana
  - Research Site, Slidell, Louisiana
  - Research Site, Auburn, Maine
  - Research Site, Bangor, Maine
  - Research Site, Baltimore, Maryland
  - Research Site, Bowie, Maryland
  - Research Site, Glen Burnie, Maryland
  - Research Site, Greenbelt, Maryland
  - Research Site, Oxon Hill, Maryland
  - Research Site, Prince Frederick, Maryland
  - Research Site, Salisbury, Maryland
  - Research Site, Haverhill, Massachusetts
  - Research Site, North Attleboro, Massachusetts
  - Research Site, Detroit, Michigan
  - Research Site, Jackson, Michigan
  - Research Site, Kalamazoo, Michigan
  - Research Site, Mount Clemens, Michigan
  - Research Site, Petoskey, Michigan
  - Research Site, Pontiac, Michigan
  - Research Site, Rochester Hills, Michigan
  - Research Site, Troy, Michigan
  - Research Site, Duluth, Minnesota
  - Research Site, Saint Paul, Minnesota
  - Research Site, Biloxi, Mississippi
  - Research Site, Jackson, Mississippi
  - Research Site, Olive Branch, Mississippi
  - Research Site, Tupelo, Mississippi
  - Research Site, Joplin, Missouri
  - Research Site, Kansas City, Missouri
  - Research Site, Lee's Summit, Missouri
  - Research Site, North Kansas City, Missouri
  - Research Site, St Louis, Missouri
  - Research Site, Helena, Montana
  - Research Site, Hastings, Nebraska
  - Research Site, Lincoln, Nebraska
  - Research Site, Las Vegas, Nevada
  - Research Site, Bridgewater, New Jersey
  - Research Site, East Brunswick, New Jersey
  - Research Site, Flemington, New Jersey
  - Research Site, Morristown, New Jersey
  - Research Site, Somerset, New Jersey
  - Research Site, Toms River, New Jersey
  - Research Site, Voorhees Township, New Jersey
  - Research Site, Albuquerque, New Mexico
  - Research Site, Albany, New York
  - Research Site, Binghamton, New York
  - Research Site, Buffalo, New York
  - Research Site, Hawthorne, New York
  - Research Site, Manhasset, New York
  - Research Site, New Windsor, New York
  - Research Site, New York, New York
  - Research Site, Orchard Park, New York
  - Research Site, Poughkeepsie, New York
  - Research Site, Saratoga Springs, New York
  - Research Site, Stony Brook, New York
  - Research Site, The Bronx, New York
  - Research Site, Utica, New York
  - Research Site, Asheville, North Carolina
  - Research Site, Calabash, North Carolina
  - Research Site, Cary, North Carolina
  - Research Site, Clayton, North Carolina
  - Research Site, High Point, North Carolina
  - Research Site, Lenoir, North Carolina
  - Research Site, Morganton, North Carolina
  - Research Site, Pinehurst, North Carolina
  - Research Site, Raleigh, North Carolina
  - Research Site, Rocky Mount, North Carolina
  - Research Site, Sanford, North Carolina
  - Research Site, Smithfield, North Carolina
  - Research Site, Tabor City, North Carolina
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Fargo, North Dakota
  - Research Site, Akron, Ohio
  - Research Site, Canton, Ohio
  - Research Site, Cincinnati, Ohio
  - Research Site, Cleveland, Ohio
  - Research Site, Dayton, Ohio
  - Research Site, Kettering, Ohio
  - Research Site, Lyndhurst, Ohio
  - Research Site, Springfield, Ohio
  - Research Site, Willoughby, Ohio
  - Research Site, Youngstown, Ohio
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Hillsboro, Oregon
  - Research Site, Medford, Oregon
  - Research Site, Butler, Pennsylvania
  - Research Site, Camp Hill, Pennsylvania
  - Research Site, Danville, Pennsylvania
  - Research Site, Doylestown, Pennsylvania
  - Research Site, Erie, Pennsylvania
  - Research Site, Harleysville, Pennsylvania
  - Research Site, Indiana, Pennsylvania
  - Research Site, Newport, Pennsylvania
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Port Matilda, Pennsylvania
  - Research Site, Scranton, Pennsylvania
  - Research Site, Wyomissing, Pennsylvania
  - Research Site, Yardley, Pennsylvania
  - Research Site, Providence, Rhode Island
  - Research Site, Columbia, South Carolina
  - Research Site, Greenwood, South Carolina
  - Research Site, North Myrtle Beach, South Carolina
  - Research Site, Rock Hill, South Carolina
  - Research Site, Simpsonville, South Carolina
  - Research Site, Varnville, South Carolina
  - Research Site, Rapid City, South Dakota
  - Research Site, Sioux Falls, South Dakota
  - Research Site, Bristol, Tennessee
  - Research Site, Jackson, Tennessee
  - Research Site, Knoxville, Tennessee
  - Research Site, Nashville, Tennessee
  - Research Site, Tullahoma, Tennessee
  - Research Site, Amarillo, Texas
  - Research Site, Arlington, Texas
  - Research Site, Austin, Texas
  - Research Site, Beaumont, Texas
  - Research Site, Channelview, Texas
  - Research Site, Dallas, Texas
  - Research Site, Fort Sam Houston, Texas
  - Research Site, Fort Worth, Texas
  - Research Site, Georgetown, Texas
  - Research Site, Houston, Texas
  - Research Site, Huntsville, Texas
  - Research Site, Katy, Texas
  - Research Site, Kingwood, Texas
  - Research Site, Lubbock, Texas
  - Research Site, McAllen, Texas
  - Research Site, Pharr, Texas
  - Research Site, Plano, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Shavano Park, Texas
  - Research Site, Bountiful, Utah
  - Research Site, Draper, Utah
  - Research Site, Salt Lake City, Utah
  - Research Site, Alexandria, Virginia
  - Research Site, Arlington, Virginia
  - Research Site, Danville, Virginia
  - Research Site, Falls Church, Virginia
  - Research Site, Manassas, Virginia
  - Research Site, Roanoke, Virginia
  - Research Site, Port Orchard, Washington
  - Research Site, Seattle, Washington
  - Research Site, Huntington, West Virginia
  - Research Site, Kenosha, Wisconsin
  - Research Site, Waukesha, Wisconsin
- Argentina (14):
  - Research Site, Buenos Aires
  - Research Site, Ciudad Autonomade Buenos Aires
  - Research Site, Ciudad Autónoma de Bs. As.
  - Research Site, Ciudadela
  - Research Site, Córdoba
  - Research Site, Mar del Plata
  - Research Site, Ranelagh
  - Research Site, Rosario
  - Research Site, San Luis
  - Research Site, San Miguel de Tucumán
  - Research Site, San Nicolás
  - Research Site, Santa Fe
  - Research Site, Venado Tuerto
  - Research Site, Villa María
- Australia (14):
  - Research Site, Adelaide
  - Research Site, Ashford
  - Research Site, Coffs Harbour
  - Research Site, Fitzroy
  - Research Site, Fullarton
  - Research Site, Geelong
  - Research Site, Heidelberg West
  - Research Site, Herston
  - Research Site, Joondalup
  - Research Site, Maroubra
  - Research Site, Melbourne
  - Research Site, Merewether
  - Research Site, Milton
  - Research Site, Murdoch
- Austria (7):
  - Research Site, Braunau am Inn
  - Research Site, Eisenstadt
  - Research Site, Feldkirch
  - Research Site, Innsbruck
  - Research Site, Saint Stefan/Stainz
  - Research Site, Salzburg
  - Research Site, Vienna
- Belgium (17):
  - Research Site, Aalst
  - Research Site, Bonheiden
  - Research Site, Bouge
  - Research Site, Bruges
  - Research Site, De Pinte
  - Research Site, Genk
  - Research Site, Ghent
  - Research Site, Hasselt
  - Research Site, Huy
  - Research Site, Leuven
  - Research Site, Liège
  - Research Site, Mechelen
  - Research Site, Mol
  - Research Site, Overpelt
  - Research Site, Roeselare
  - Research Site, Yvoir
  - Research Site, Zottegem
- Brazil (23):
  - Research Site, Belo Horizonte
  - Research Site, Blumenau
  - Research Site, Brasillia
  - Research Site, Brasília
  - Research Site, Campina Grande do Sul
  - Research Site, Campinas
  - Research Site, Campo Grande
  - Research Site, Cariacica
  - Research Site, Curitiba
  - Research Site, Fortaleza
  - Research Site, Goiânia
  - Research Site, Maringá
  - Research Site, Marília
  - Research Site, Porto Alegre
  - Research Site, Ribeirão Preto
  - Research Site, Rio de Janeiro
  - Research Site, S.J.Rio Preto
  - Research Site, São José dos Campos
  - Research Site, São Paulo
  - Research Site, Tatuí
  - Research Site, Uberlândia
  - Research Site, Vitória
  - Research Site, Votuporanga
- Bulgaria (21):
  - Research Site, Blagoevgrad
  - Research Site, Botevgrad
  - Research Site, Burgas
  - Research Site, Dimitrovgrad
  - Research Site, Dupnitsa
  - Research Site, Gabrovo
  - Research Site, Haskovo
  - Research Site, Kozloduy
  - Research Site, Kyustendil
  - Research Site, Lom
  - Research Site, Pazardzhik
  - Research Site, Pleven
  - Research Site, Plovdiv
  - Research Site, Rousse
  - Research Site, Sandanski
  - Research Site, Sevlievo
  - Research Site, Sliven
  - Research Site, Sofia
  - Research Site, Stara Zagora
  - Research Site, Varna
  - Research Site, Yambol
- Canada (44):
  - Research Site, Calgary, Alberta
  - Research Site, Edmonton, Alberta
  - Research Site, Red Deer, Alberta
  - Research Site, Spruce Grove, Alberta
  - Research Site, Kelowna, British Columbia
  - Research Site, New Westminster, British Columbia
  - Research Site, Penticton, British Columbia
  - Research Site, Surrey, British Columbia
  - Research Site, Vancouver, British Columbia
  - Research Site, Victoria, British Columbia
  - Research Site, Saint John, New Brunswick
  - Research Site, Mount Pearl, Newfoundland and Labrador
  - Research Site, St. John's, Newfoundland and Labrador
  - Research Site, Halifax, Nova Scotia
  - Research Site, Brampton, Ontario
  - Research Site, Cambridge, Ontario
  - Research Site, Cornwall, Ontario
  - Research Site, Greater Sudbury, Ontario
  - Research Site, Hamilton, Ontario
  - Research Site, Jarvis, Ontario
  - Research Site, London, Ontario
  - Research Site, Newmarket, Ontario
  - Research Site, North York, Ontario
  - Research Site, Oshawa, Ontario
  - Research Site, Ottawa, Ontario
  - Research Site, Sarnia, Ontario
  - Research Site, Scarborough Village, Ontario
  - Research Site, Thornhill, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Waterloo, Ontario
  - Research Site, Brossard, Quebec
  - Research Site, Chicoutimi, Quebec
  - Research Site, Greenfield Park, Quebec
  - Research Site, Laval, Quebec
  - Research Site, Longueuil, Quebec
  - Research Site, Montreal, Quebec
  - Research Site, Québec, Quebec
  - Research Site, Saint-Charles-Borromée, Quebec
  - Research Site, Saint-Georges, Quebec
  - Research Site, Saint-Jean-sur-Richelieu, Quebec
  - Research Site, Saint-Lambert, Quebec
  - Research Site, Terrebonne, Quebec
  - Research Site, Regina, Saskatchewan
  - Research Site, Chicoutimi
- Chile (7):
  - Research Site, Concepción
  - Research Site, Los Ángeles
  - Research Site, Osorno
  - Research Site, Santiago
  - Research Site, Talcahuano
  - Research Site, Temuco
  - Research Site, Viña del Mar
- China (17):
  - Research Site, Beijing
  - Research Site, Bengbu
  - Research Site, Cangzhou
  - Research Site, Chengdu
  - Research Site, Fuzhou
  - Research Site, Guangzhou
  - Research Site, Jinan
  - Research Site, Nanchang
  - Research Site, Nanjing
  - Research Site, Pingxiang
  - Research Site, Shanghai
  - Research Site, Shenyang
  - Research Site, Taiyuan
  - Research Site, Tianjin
  - Research Site, Wuhan
  - Research Site, Xi'an
  - Research Site, Yinchuan
- Colombia (9):
  - Research Site, Armenia
  - Research Site, Barranquilla
  - Research Site, Bogotá
  - Research Site, Bucaramanga
  - Research Site, Cali
  - Research Site, Cartagena
  - Research Site, Floridablanca
  - Research Site, Manizales
  - Research Site, Medellín
- Czechia (22):
  - Research Site, Benešov
  - Research Site, Brno
  - Research Site, Chomutov
  - Research Site, Česká Lípa
  - Research Site, Frýdek-Místek
  - Research Site, Jablonec nad Nisou
  - Research Site, Karlovy Vary
  - Research Site, Kolín
  - Research Site, Kutná Hora
  - Research Site, Louny
  - Research Site, Olomouc
  - Research Site, Ostrava
  - Research Site, Ostrava-Dubina
  - Research Site, Pelhřimov
  - Research Site, Prague
  - Research Site, Pribram VIII
  - Research Site, Slaný
  - Research Site, Třebíč
  - Research Site, Turnov
  - Research Site, Ústí nad Labem
  - Research Site, Ústí nad Orlicí
  - Research Site, Zábřeh nad Odrou
- Denmark (13):
  - Research Site, Aarhus N
  - Research Site, Esbjerg
  - Research Site, Hjørring
  - Research Site, Hvidovre
  - Research Site, Kolding
  - Research Site, Købehhavn Ø
  - Research Site, København NV
  - Research Site, Næstved
  - Research Site, Odense C
  - Research Site, Roslev
  - Research Site, Svendborg
  - Research Site, Viborg
  - Research Site, Værløse
- Finland (9):
  - Research Site, Helsinki
  - Research Site, Joensuu
  - Research Site, Jyväskylä
  - Research Site, Kokkola
  - Research Site, Kuopio
  - Research Site, Lahti
  - Research Site, Oulu
  - Research Site, Tampere
  - Research Site, Turku
- France (15):
  - Research Site, Avignon
  - Research Site, Bayonne
  - Research Site, Bobigny
  - Research Site, Corbeil-Essonnes
  - Research Site, Dijon
  - Research Site, La Rochelle
  - Research Site, Le Coudray
  - Research Site, Lyon
  - Research Site, Montauban
  - Research Site, Nice
  - Research Site, Nîmes
  - Research Site, Paris
  - Research Site, Toulouse
  - Research Site, Tourcoing
  - Research Site, Tours
- Germany (19):
  - Research Site, Altdorf
  - Research Site, Aschaffenburg
  - Research Site, Bad Krozingen
  - Research Site, Berlin
  - Research Site, Cologne
  - Research Site, Dresden
  - Research Site, Hamburg
  - Research Site, Kassel
  - Research Site, Leipzig
  - Research Site, Markkleeberg
  - Research Site, Meißen
  - Research Site, Mühldorf
  - Research Site, München
  - Research Site, Neuwied
  - Research Site, Nuremberg
  - Research Site, Papenburg
  - Research Site, Schwerin
  - Research Site, Wangen
  - Research Site, Wermsdorf
- Research Site, Hong Kong, Hong Kong
- Hungary (19):
  - Research Site, Balatonfüred
  - Research Site, Berettyóújfalu
  - Research Site, Budapest
  - Research Site, Debrecen
  - Research Site, Eger
  - Research Site, Hajdúszoboszló
  - Research Site, Kalocsa
  - Research Site, Kecskemét
  - Research Site, Kistarcsa
  - Research Site, Kisvárda
  - Research Site, Mosonmagyaróvár
  - Research Site, Nyíregyháza
  - Research Site, Pásztó
  - Research Site, Pécs
  - Research Site, Sopron
  - Research Site, Szentes
  - Research Site, Székesfehérvár
  - Research Site, Szolnok
  - Research Site, Zalaegerszeg
- India (6):
  - Research Site, Ahmedabad
  - Research Site, Bangalore
  - Research Site, Chennai
  - Research Site, Kolkata
  - Research Site, New Delhi
  - Research Site, Pune
- Israel (6):
  - Research Site, Haifa
  - Research Site, Holon
  - Research Site, Jerusalem
  - Research Site, Nahariya
  - Research Site, Petah Tikva
  - Research Site, Tel Aviv
- Italy (14):
  - Research Site, Bari
  - Research Site, Bergamo
  - Research Site, Bologna
  - Research Site, Florence
  - Research Site, Genova
  - Research Site, Milan
  - Research Site, Napoli
  - Research Site, Novara
  - Research Site, Pavia
  - Research Site, Rivoli
  - Research Site, Roma
  - Research Site, San Giovanni Rotondo
  - Research Site, Udine
  - Research Site, Viterbo
- Japan (47):
  - Research Site, Adachi-ku
  - Research Site, Beppu-shi
  - Research Site, Chikushino-shi
  - Research Site, Chūōku
  - Research Site, Daito-shi
  - Research Site, Edogawa-ku
  - Research Site, Fujisawa-shi
  - Research Site, Fukui-shi
  - Research Site, Fukuoka
  - Research Site, Funabashi-shi
  - Research Site, Fussa-shi
  - Research Site, Gifu
  - Research Site, Hachioji-shi
  - Research Site, Hitachi-shi
  - Research Site, Isehara-shi
  - Research Site, Iwakuni-shi
  - Research Site, Kagoshima
  - Research Site, Kawanishi-shi
  - Research Site, Kishiwada-shi
  - Research Site, Kobe
  - Research Site, Koga-shi
  - Research Site, Koriyama-shi
  - Research Site, Kumamoto
  - Research Site, Kure-shi
  - Research Site, Kurume-shi
  - Research Site, Kyoto
  - Research Site, Matsudo-shi
  - Research Site, Miura-gun
  - Research Site, Okayama
  - Research Site, Osaka
  - Research Site, Otaru-shi
  - Research Site, Sanyoonoda-shi
  - Research Site, Sapporo
  - Research Site, Sayama-shi
  - Research Site, Shimajiri-gun
  - Research Site, Takamatsu
  - Research Site, Takasaki-shi
  - Research Site, Takayama-shi
  - Research Site, Toyohashi
  - Research Site, Toyota-shi
  - Research Site, Tsuchiura-shi
  - Research Site, Uji-shi
  - Research Site, Urasoe-shi
  - Research Site, Ureshino-shi
  - Research Site, Wakayama
  - Research Site, Wako-shi
  - Research Site, Yokohama
- Mexico (12):
  - Research Site, Culiacán
  - Research Site, D.F
  - Research Site, Guadalajara
  - Research Site, México
  - Research Site, Monterrey
  - Research Site, Morelia
  - Research Site, Nuevo León
  - Research Site, Pachuca
  - Research Site, Querétaro
  - Research Site, Tijuana
  - Research Site, Xalapa
  - Research Site, Zapopan
- Netherlands (23):
  - Research Site, 's-Hertogenbosch
  - Research Site, Alkmaar
  - Research Site, Amsterdam
  - Research Site, Arnhem
  - Research Site, Beverwijk
  - Research Site, Blaricum
  - Research Site, Breda
  - Research Site, Delft
  - Research Site, Eindhoven
  - Research Site, Emmen
  - Research Site, Enschede
  - Research Site, Goes
  - Research Site, Helmond
  - Research Site, Hoofddorp
  - Research Site, Hoogeveen
  - Research Site, Maastricht
  - Research Site, Roosendaal
  - Research Site, Rotterdam
  - Research Site, Schiedam
  - Research Site, Stadskanaal
  - Research Site, Tiel
  - Research Site, Uden
  - Research Site, Veldhoven
- Norway (13):
  - Research Site, Ålesund
  - Research Site, Bergen
  - Research Site, Bodø
  - Research Site, Kongsvinger
  - Research Site, Lillehammer
  - Research Site, Oslo
  - Research Site, Sandefjord
  - Research Site, Skedsmokorset
  - Research Site, Skien
  - Research Site, Stavanger
  - Research Site, Svelvik
  - Research Site, Tromsø
  - Research Site, Trondheim
- Peru (5):
  - Research Site, Arequipa
  - Research Site, Callao
  - Research Site, Chiclayo
  - Research Site, Lima
  - Research Site, Miraflores
- Philippines (6):
  - Research Site, Cebu
  - Research Site, Cebu City
  - Research Site, City of Taguig
  - Research Site, Davao City
  - Research Site, Pasig
  - Research Site, Quezon City
- Poland (55):
  - Research Site, Bialystok
  - Research Site, Biała Rawska
  - Research Site, Bielsko-Biala
  - Research Site, Bochnia
  - Research Site, Bydgoszcz
  - Research Site, Chojnice
  - Research Site, Chorzów
  - Research Site, Chrzanów
  - Research Site, Elblag
  - Research Site, Gdansk
  - Research Site, Gdynia
  - Research Site, Giżycko
  - Research Site, Grodzisk Mazowiecki
  - Research Site, Jasło
  - Research Site, Katowice
  - Research Site, Kędzierzyn-Koźle
  - Research Site, Kielce
  - Research Site, Koszalin
  - Research Site, Kościan
  - Research Site, Krakow
  - Research Site, Legnica
  - Research Site, Lodz
  - Research Site, Lubin
  - Research Site, Lublin
  - Research Site, Mikołów
  - Research Site, Myszków
  - Research Site, Nakło nad Notecią
  - Research Site, Nowogard
  - Research Site, Nysa
  - Research Site, Opole
  - Research Site, Ostrów Mazowiecka
  - Research Site, Oświęcim
  - Research Site, Poznan
  - Research Site, Puławy
  - Research Site, Płock
  - Research Site, Ruda Śląska
  - Research Site, Rzeszów
  - Research Site, Siedlce
  - Research Site, Sobótka
  - Research Site, Sokółka
  - Research Site, Staszów
  - Research Site, Szczecin
  - Research Site, Tarnów
  - Research Site, Torun
  - Research Site, Tychy
  - Research Site, Ustroń
  - Research Site, Warsaw
  - Research Site, Wierzchosławice
  - Research Site, Wroclaw
  - Research Site, Włocławek
  - Research Site, Zabrze
  - Research Site, Zamość
  - Research Site, Zgierz
  - Research Site, Zielona Góra
  - Research Site, Żnin
- Puerto Rico (2):
  - Research Site, Canovanas
  - Research Site, Cidra
- Romania (6):
  - Research Site, Bacau
  - Research Site, Bucharest
  - Research Site, Craiova
  - Research Site, Iași
  - Research Site, Piteşti
  - Research Site, Suceava
- Russia (27):
  - Research Site, Arkhangelsk
  - Research Site, Gatchina
  - Research Site, Ivanovo
  - Research Site, Izhevsk
  - Research Site, Kaluga
  - Research Site, Kazan'
  - Research Site, Kemerovo
  - Research Site, Khanty-Mansiysk
  - Research Site, Krasnodar
  - Research Site, Moscow
  - Research Site, Nizhny Novgorod
  - Research Site, Novosibirsk
  - Research Site, Omsk
  - Research Site, Perm
  - Research Site, Rostov-on-Don
  - Research Site, Ryazan
  - Research Site, Saint Petersburg
  - Research Site, Saratov
  - Research Site, StPetersburg
  - Research Site, Tomsk
  - Research Site, Tver'
  - Research Site, Tyumen
  - Research Site, Ufa
  - Research Site, Vladimir
  - Research Site, Volgograd
  - Research Site, Yaroslavl
  - Research Site, Yekaterinburg
- Saudi Arabia (4):
  - Research Site, Dammam
  - Research Site, Jeddah
  - Research Site, Khobar
  - Research Site, Riyadh
- Slovakia (14):
  - Research Site, Banská Bystrica
  - Research Site, Bratislava
  - Research Site, Brezno
  - Research Site, Košice
  - Research Site, Kráľovský Chlmec
  - Research Site, Liptovský Mikuláš
  - Research Site, Lučenec
  - Research Site, Martin
  - Research Site, Nitra
  - Research Site, Prešov
  - Research Site, Ružomberok
  - Research Site, Svidník
  - Research Site, Trnava
  - Research Site, Žilina
- South Africa (13):
  - Research Site, Alberton
  - Research Site, Benoni
  - Research Site, Bloemfontein
  - Research Site, Cape Town
  - Research Site, Durban
  - Research Site, Greenbury, Phoenix
  - Research Site, Johannesburg
  - Research Site, KwaDukuza
  - Research Site, Paarl
  - Research Site, Port Elizabeth
  - Research Site, Soweto
  - Research Site, Verulam
  - Research Site, Worcester
- South Korea (17):
  - Research Site, Anyang-si
  - Research Site, Bucheon-si
  - Research Site, Busan
  - Research Site, Changwon-si
  - Research Site, Cheonan-si
  - Research Site, Cheongju-si
  - Research Site, Daegu
  - Research Site, Daejeon
  - Research Site, Gwangju
  - Research Site, Iksan-si
  - Research Site, Incheon
  - Research Site, Jeonju
  - Research Site, Jinju
  - Research Site, Seongnam-si
  - Research Site, Seoul
  - Research Site, Suwon
  - Research Site, Wŏnju
- Spain (27):
  - Research Site, A Coruña
  - Research Site, Alcalá de Henares
  - Research Site, Alicante
  - Research Site, Barcelona
  - Research Site, Bilbao
  - Research Site, Cáceres
  - Research Site, El Palmar
  - Research Site, Ferrol (A Coruña)
  - Research Site, Girona
  - Research Site, Granada
  - Research Site, Huelva
  - Research Site, L'Hospitalet de Llobregat
  - Research Site, La Laguna (Tenerife)
  - Research Site, Madrid
  - Research Site, Majadahonda
  - Research Site, Málaga
  - Research Site, Móstoles
  - Research Site, Pontevedra
  - Research Site, Sabadell
  - Research Site, San Sebastián de los Reyes
  - Research Site, Sant Joan d'Alacant
  - Research Site, Santander
  - Research Site, Santiago(A Coruña)
  - Research Site, Seville
  - Research Site, Son Ferriol
  - Research Site, Valdemoro
  - Research Site, Valencia
- Sweden (10):
  - Research Site, Gothenburg
  - Research Site, Jönköping
  - Research Site, Lessebo
  - Research Site, Lund
  - Research Site, Malmo
  - Research Site, Örebro
  - Research Site, Rättvik
  - Research Site, Stockholm
  - Research Site, Uppsala
  - Research Site, Västerås
- Taiwan (10):
  - Research Site, Changhua
  - Research Site, Hsinchu
  - Research Site, Hualien City
  - Research Site, Kaohsiung City
  - Research Site, Kweishan Shiang
  - Research Site, New Taipei City
  - Research Site, Pingtung City
  - Research Site, Taichung
  - Research Site, Tainan
  - Research Site, Taipei
- Thailand (6):
  - Research Site, Bangkok
  - Research Site, Bangkoknoi
  - Research Site, Chiang Mai
  - Research Site, Hat Yai
  - Research Site, Muang
  - Research Site, Naimuang
- Turkey (Türkiye) (6):
  - Research Site, Adana
  - Research Site, Ankara
  - Research Site, Antalya
  - Research Site, Aydin
  - Research Site, Istanbul
  - Research Site, Mersin
- Ukraine (16):
  - Research Site, Belo Horizonte
  - Research Site, Cherkasy
  - Research Site, Dnipro
  - Research Site, Ivano-Frankivsk
  - Research Site, Kharkiv Region
  - Research Site, Kyiv
  - Research Site, Lutsk
  - Research Site, Lviv
  - Research Site, Mykolaiv
  - Research Site, Odesa
  - Research Site, Poltava
  - Research Site, Rivne
  - Research Site, Ternopil
  - Research Site, Uzhhorod
  - Research Site, Vinnytsia
  - Research Site, Zaporizhzhia
- United Kingdom (27):
  - Research Site, Airdrie
  - Research Site, Antrim
  - Research Site, Belfast
  - Research Site, Chesterfield
  - Research Site, Coventry
  - Research Site, Doncaster
  - Research Site, Dundee
  - Research Site, Durham
  - Research Site, Exeter
  - Research Site, Faringdon
  - Research Site, Glasgow
  - Research Site, Harrogate
  - Research Site, High Wycombe
  - Research Site, London
  - Research Site, Middlesbrough
  - Research Site, Newcastle upon Tyne
  - Research Site, Northampton
  - Research Site, Nottingham
  - Research Site, Paisley
  - Research Site, Peterborough
  - Research Site, Plymouth
  - Research Site, Rotherham
  - Research Site, Rothwell
  - Research Site, Sheffield
  - Research Site, Swansea
  - Research Site, Torquay
  - Research Site, York
- Vietnam (3):
  - Research Site, Hanoi
  - Research Site, Ho Chi Minh City
  - Research Site, Hochiminh

REFERENCES:
- [Background] Steg PG, Bhatt DL, Simon T, Fox K, Mehta SR, Harrington RA, Held C, Andersson M, Himmelmann A, Ridderstrale W, Leonsson-Zachrisson M, Liu Y, Opolski G, Zateyshchikov D, Ge J, Nicolau JC, Corbalan R, Cornel JH, Widimsky P, Leiter LA; THEMIS Steering Committee and Investigators. Ticagrelor in Patients with Stable Coronary Disease and Diabetes. N Engl J Med. 2019 Oct 3;381(14):1309-1320. doi: 10.1056/NEJMoa1908077. Epub 2019 Sep 1. PMID 31475798
- [Background] Bhatt DL, Steg PG, Mehta SR, Leiter LA, Simon T, Fox K, Held C, Andersson M, Himmelmann A, Ridderstrale W, Chen J, Song Y, Diaz R, Goto S, James SK, Ray KK, Parkhomenko AN, Kosiborod MN, McGuire DK, Harrington RA; THEMIS Steering Committee and Investigators. Ticagrelor in patients with diabetes and stable coronary artery disease with a history of previous percutaneous coronary intervention (THEMIS-PCI): a phase 3, placebo-controlled, randomised trial. Lancet. 2019 Sep 28;394(10204):1169-1180. doi: 10.1016/S0140-6736(19)31887-2. Epub 2019 Sep 1. PMID 31484629
- [Background] Bhatt DL, Fox K, Harrington RA, Leiter LA, Mehta SR, Simon T, Andersson M, Himmelmann A, Ridderstrale W, Held C, Steg PG; THEMIS Steering Committee. Rationale, design and baseline characteristics of the effect of ticagrelor on health outcomes in diabetes mellitus patients Intervention study. Clin Cardiol. 2019 May;42(5):498-505. doi: 10.1002/clc.23164. Epub 2019 Apr 9. PMID 30788847
- [Derived] Bonaca MP, Bhatt DL, Simon T, Fox KM, Mehta S, Harrington RA, Leiter LA, Capell WH, Held C, Himmelmann A, Ridderstrale W, Chen J, Lee JJ, Song Y, Andersson M, Prats J, Kosiborod M, McGuire DK, Steg PG. Limb Outcomes With Ticagrelor Plus Aspirin in Patients With Diabetes Mellitus and Atherosclerosis. J Am Coll Cardiol. 2024 Apr 30;83(17):1627-1636. doi: 10.1016/j.jacc.2024.03.377. PMID 38658101
- [Derived] Abtan J, Bhatt DL, Elbez Y, Ducrocq G, Goto S, Smith SC Jr, Ohman EM, Eagle KA, Fox K, Harrington RA, Leiter LA, Mehta SR, Simon T, Petrov I, Sinnaeve PR, Pais P, Lev E, Bueno H, Wilson P, Steg PG; REACH Registry Investigators. External applicability of the Effect of ticagrelor on Health Outcomes in diabEtes Mellitus patients Intervention Study (THEMIS) trial: An analysis of patients with diabetes and coronary artery disease in the REduction of Atherothrombosis for Continued Health (REACH) registry. Int J Cardiol. 2023 Jan 1;370:51-57. doi: 10.1016/j.ijcard.2022.10.132. Epub 2022 Oct 19. PMID 36270493
- [Derived] Wittbrodt E, Bhalla N, Sundell KA, Hunt P, Wong ND, Kuster M, Mellstrom C. Assessment of The High risk and unmEt Need in patients with CAD and type 2 diabetes (ATHENA): US healthcare resource use, cost, and burden of illness in a commercially insured population. J Diabetes Complications. 2021 Apr;35(4):107859. doi: 10.1016/j.jdiacomp.2021.107859. Epub 2021 Jan 20. PMID 33558152
- [Derived] Held P, Himmelmann A, Ditmarsch M. Ticagrelor for the treatment of atherosclerotic disease: insights from the PARTHENON clinical development program. Future Cardiol. 2016 Jul;12(4):405-18. doi: 10.2217/fca-2016-0028. Epub 2016 May 10. PMID 27160944
- See also: D513BC00001_CSP_redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D513BC00001&attachmentIdentifier=04c28e5e-3d5e-4b76-824f-220474f85319&fileName=D513BC00001_CSP_redacted.pdf&versionIdentifier=
- See also: D513BC00001_SAP_redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D513BC00001&attachmentIdentifier=40d0421c-d5ae-4781-a3f8-69e550dcfd03&fileName=D513BC00001_SAP_redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 1315 study sites in 42 countries enrolled patients. The first patient was enrolled on 10 February 2014. The last patient visit took place on 25 January 2019.
Pre-assignment Details: Enrolled patients randomised to study drug 95.8%; n =19271, of which 51 patients were randomised to study drug at a site prematurely closed by sponsor and excluded from the study results. Patients who were not randomised 4.2%; n=837. Patient did not meet inclusion/exclusion criteria n=454, Patient decision n=256, Death n=1, Other reason n=131.
Period: Overall Study
Arm/Group | Ticagrelor 60 mg | Ticagrelor Placebo
Started (Includes patients that were randomised to study drug) | 9645 | 9626
Completed (Patients who did not withdrew informed consent, were not LTFU and not excluded from the analyses) | 9496 | 9503
Not Completed | 149 | 123
Not completed — Lost to Follow-up | 6 | 4
Not completed — Withdrawal by Subject | 117 | 94
Not completed — Site prematurely closed by sponsor | 26 | 25

BASELINE CHARACTERISTICS:
Population: Of the 19271 patients randomised to study drug, 51 patients were randomised to study drug at a site prematurely closed by sponsor and excluded from the study results. 19220 were included in the evaluation of study results.
Groups:
- Total: Total of all reporting groups
Arm/Group | Ticagrelor 60 mg | Ticagrelor Placebo | Total
Number analyzed (Participants) | 9619 | 9601 | 19220
Age, Continuous [Mean (Standard Deviation); unit: Years] | 66.3 (7.8) | 66.3 (7.7) | 66.3 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3043 | 2988 | 6031
  Male | 6576 | 6613 | 13189
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 6838 | 6858 | 13696
  Black or african american | 205 | 198 | 403
  Asian | 2211 | 2195 | 4406
  Native hawaiian or other pacific islander | 7 | 7 | 14
  American indian or alaska native | 161 | 152 | 313
  Other | 197 | 191 | 388
Region of Enrollment [Number; unit: Participants]
  USA | 1126 | 1140 | 2266
  Argentina | 195 | 199 | 394
  Australia | 94 | 94 | 188
  Austria | 42 | 45 | 87
  Belgium | 109 | 108 | 217
  Bulgaria | 435 | 443 | 878
  Brazil | 412 | 399 | 811
  Canada | 364 | 365 | 729
  Chile | 152 | 148 | 300
  China | 456 | 454 | 910
  Colombia | 68 | 68 | 136
  Czech Republic | 304 | 298 | 602
  Germany | 277 | 270 | 547
  Denmark | 123 | 120 | 243
  Spain | 170 | 170 | 340
  Finland | 60 | 58 | 118
  France | 85 | 87 | 172
  United Kingdom | 123 | 123 | 246
  Hong Kong | 76 | 76 | 152
  Hungary | 306 | 310 | 616
  India | 147 | 145 | 292
  Israel | 60 | 57 | 117
  Italy | 67 | 63 | 130
  Japan | 246 | 250 | 496
  Korea, Republic Of | 433 | 437 | 870
  Mexico | 182 | 182 | 364
  Netherlands | 242 | 237 | 479
  Norway | 95 | 96 | 191
  Peru | 91 | 82 | 173
  Philippines | 47 | 45 | 92
  Poland | 815 | 821 | 1636
  Romania | 37 | 43 | 80
  Russia | 561 | 560 | 1121
  Saudi Arabia | 79 | 76 | 155
  Slovakia | 122 | 122 | 244
  Sweden | 110 | 114 | 224
  Thailand | 115 | 116 | 231
  Turkey | 113 | 112 | 225
  Taiwan, Province Of China | 402 | 401 | 803
  Ukraine | 399 | 393 | 792
  Viet Nam | 129 | 125 | 254
  South Africa | 150 | 149 | 299

OUTCOME MEASURES:

1. Primary Outcome: Composite of Cardiovascular (CV) Death, MI or Stroke
Description: Participants with Cardiovascular (CV) death, myocardial infarction (MI) or stroke. If no event, censoring occurs at the earliest of PACD, last endpoint assessment date and non-CV death date.
Time Frame: From randomisation to primary analysis censoring date (PACD). Median time in study until PACD was 40 months.
Population: The population was the full analysis set, which included all randomised patients except the 51 patients who were randomised to study drug at a site prematurely closed by sponsor.
Measure: Number; unit: Number of participants with event
Arm/Group | Ticagrelor 60 mg | Ticagrelor Placebo
Number analyzed (Participants) | 9619 | 9601
Number of participants with event | 736 | 818
Statistical Analysis 1: Comparison: Ticagrelor 60 mg vs Ticagrelor Placebo; Test type: Superiority; p = 0.0378, Regression, Cox — The hypothesis will be tested at the 4.96% two-sided significance level to account for the planned interim analysis with the overall type I error preserved at 5%. A hierarchical test sequence will be used to address the issue of multiple testing; Hazard Ratio (HR) = 0.90, 95% CI 2-sided [0.81 to 0.99]

2. Secondary Outcome: CV Death
Description: Participants with Cardiovascular (CV) death. If no event, censoring occurs at the earliest of PACD, last endpoint assessment date and non-CV death date.
Time Frame: From randomisation to primary analysis censoring date (PACD). Median time in study until PACD was 40 months.
Population: as for outcome 1
Measure: Number; unit: Number of participants with event
Arm/Group | Ticagrelor 60 mg | Ticagrelor Placebo
Number analyzed (Participants) | 9619 | 9601
Number of participants with event | 364 | 357
Statistical Analysis 1: Comparison: Ticagrelor 60 mg vs Ticagrelor Placebo; Test type: Superiority; p = 0.7883, Regression, Cox — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 1.02, 95% CI 2-sided [0.88 to 1.18]

3. Secondary Outcome: MI
Description: Participants with myocardial infarction. If no event, censoring occurs at the earliest of primary analysis censoring date (PACD), last endpoint assessment date and death date
Time Frame: From randomisation to primary analysis censoring date (PACD). Median time in study until PACD was 40 months.
Population: as for outcome 1
Measure: Number; unit: Number of participants with event
Arm/Group | Ticagrelor 60 mg | Ticagrelor Placebo
Number analyzed (Participants) | 9619 | 9601
Number of participants with event | 274 | 328
Statistical Analysis 1: Comparison: Ticagrelor 60 mg vs Ticagrelor Placebo; Test type: Superiority; p = 0.0294, Regression, Cox — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.84, 95% CI 2-sided [0.71 to 0.98]

4. Secondary Outcome: Ischaemic Stroke
Description: Participants with ischaemic stroke. If no event, censoring occurs at the earliest of PACD, last endpoint assessment date and death date.
Time Frame: From randomisation to primary analysis censoring date (PACD). Median time in study until PACD was 40 months.
Population: as for outcome 1
Measure: Number; unit: Number of participants with event
Arm/Group | Ticagrelor 60 mg | Ticagrelor Placebo
Number analyzed (Participants) | 9619 | 9601
Number of participants with event | 152 | 191
Statistical Analysis 1: Comparison: Ticagrelor 60 mg vs Ticagrelor Placebo; Test type: Superiority; p = 0.0375, Regression, Cox — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.80, 95% CI 2-sided [0.64 to 0.99]

5. Secondary Outcome: All-cause Death
Description: Participants with all-cause death. If no event, censoring occurs at the earliest of PACD and last endpoint assessment date. Includes deaths based on publically available vital status data in patients who have withdrawn consent.
Time Frame: From randomisation to primary analysis censoring date (PACD). Median time in study until PACD was 40 months.
Population: as for outcome 1
Measure: Number; unit: Number of participants with event
Arm/Group | Ticagrelor 60 mg | Ticagrelor Placebo
Number analyzed (Participants) | 9619 | 9601
Number of participants with event | 579 | 592
Statistical Analysis 1: Comparison: Ticagrelor 60 mg vs Ticagrelor Placebo; Test type: Superiority; p = 0.6846, Regression, Cox; Hazard Ratio (HR) = 0.98, 95% CI 2-sided [0.87 to 1.10]

6. Other Pre Specified Outcome: TIMI Major Bleeding Event (Primary Safety Objective)
Description: Participants with TIMI major bleeding event. If no event, censoring occurs at the earliest of last endpoint assessment date, death date and 7 days following the date of last dose of study medication
Time Frame: From randomisation to 7 days following the date of last dose of study medication. Maximum duration of exposure was 59 months.
Population: The population was the safety analysis set, which included all patients who received at least 1 dose of randomised ticagrelor or placebo
Measure: Number; unit: Number of participants with event
Arm/Group | Ticagrelor 60 mg | Ticagrelor Placebo
Number analyzed (Participants) | 9562 | 9531
Number of participants with event | 206 | 100
Statistical Analysis 1: Comparison: Ticagrelor 60 mg vs Ticagrelor Placebo; Test type: Superiority; p < 0.0001, Regression, Cox; Hazard Ratio (HR) = 2.32, 95% CI 2-sided [1.82 to 2.94]

7. Other Pre Specified Outcome: TIMI Major or Minor Bleeding Event
Description: Participants with TIMI major or minor bleeding event. If no event, censoring occurs at the earliest of last endpoint assessment date, death date and 7 days following the date of last dose of study medication
Time Frame: as for outcome 6
Population: as for outcome 6
Measure: Number; unit: Number of participants with event
Arm/Group | Ticagrelor 60 mg | Ticagrelor Placebo
Number analyzed (Participants) | 9562 | 9531
Number of participants with event | 285 | 129
Statistical Analysis 1: Comparison: Ticagrelor 60 mg vs Ticagrelor Placebo; Test type: Superiority; p < 0.0001, Regression, Cox; Hazard Ratio (HR) = 2.49, 95% CI 2-sided [2.02 to 3.07]

8. Other Pre Specified Outcome: PLATO Major Bleeding Event
Description: Participants with PLATO major bleeding event. If no event, censoring occurs at the earliest of last endpoint assessment date, death date and 7 days following the date of last dose of study medication
Time Frame: as for outcome 6
Population: as for outcome 6
Measure: Number; unit: Number of participants with event
Arm/Group | Ticagrelor 60 mg | Ticagrelor Placebo
Number analyzed (Participants) | 9562 | 9531
Number of participants with event | 310 | 145
Statistical Analysis 1: Comparison: Ticagrelor 60 mg vs Ticagrelor Placebo; Test type: Superiority; p < 0.0001, Regression, Cox; Hazard Ratio (HR) = 2.41, 95% CI 2-sided [1.98 to 2.93]

9. Other Pre Specified Outcome: Permanent Discontinuation of Study Medication Due to Any Bleeding Event
Description: Participants with permanent discontinuation of study medication due to any bleeding event. If no event, censoring occurs at the earliest of last endpoint assessment date, death date and the date of last dose of study medication
Time Frame: as for outcome 6
Population: as for outcome 6
Measure: Number; unit: Number of participants with event
Arm/Group | Ticagrelor 60 mg | Ticagrelor Placebo
Number analyzed (Participants) | 9562 | 9531
Number of participants with event | 466 | 125
Statistical Analysis 1: Comparison: Ticagrelor 60 mg vs Ticagrelor Placebo; Test type: Superiority; p < 0.0001, Regression, Cox; Hazard Ratio (HR) = 4.04, 95% CI 2-sided [3.32 to 4.92]

ADVERSE EVENTS:
Time Frame: All-cause death includes all deaths that occur between randomisation and last visit (before and after primary analysis censoring date, and including vital status known from public records). The other adverse event categories are presented with event onset date between randomisation to 7 days following the date of last dose of study medication. Maximum duration of exposure was 59 months.
Description: All-cause death was assessed for all randomised participants, except the 51 patients who were randomised to study drug at a site prematurely closed by sponsor.
  Systematic assessment of suspected bleeding events, suspected endpoint events, SAEs, AEs that leads to permanent discontinuation of study drug and non-serious AEs of interest. The analysis set included all patients who received at least 1 dose of study drug, except those patients randomised at the prematurely closed site.
Arm/Group | Ticagrelor 60 mg | Ticagrelor Placebo
All-Cause Mortality (participants affected / at risk) | 589/9619 | 602/9601
Serious Adverse Events (participants affected / at risk) | 3049/9562 | 3210/9531
Other Adverse Events (participants affected / at risk) | 1951/9562 | 610/9531
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ticagrelor 60 mg (N=9562) | Ticagrelor Placebo (N=9531)
Abdominal lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Agranulocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 20 (20) | 14 (14)
Anaemia macrocytic (Blood and lymphatic system disorders) | 3 (3) | 0 (0)
Anaemia of chronic disease (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Anaemia of malignant disease (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Anaemia vitamin b12 deficiency (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Deficiency anaemia (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 10 (10) | 3 (3)
Hypochromic anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Immune thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Increased tendency to bruise (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 26 (26) | 6 (6)
Leukocytosis (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Microcytic anaemia (Blood and lymphatic system disorders) | 3 (3) | 1 (1)
Nephrogenic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Normocytic anaemia (Blood and lymphatic system disorders) | 2 (3) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 3 (3) | 0 (0)
Splenic infarction (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Spontaneous haematoma (Blood and lymphatic system disorders) | 3 (3) | 2 (2)
Spontaneous haemorrhage (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 20 (20) | 22 (22)
Acute left ventricular failure (Cardiac disorders) | 5 (6) | 2 (2)
Acute myocardial infarction (Cardiac disorders) | 126 (133) | 197 (203)
Adams-stokes syndrome (Cardiac disorders) | 2 (2) | 0 (0)
Angina pectoris (Cardiac disorders) | 200 (239) | 251 (267)
Angina unstable (Cardiac disorders) | 354 (403) | 405 (449)
Aortic valve disease (Cardiac disorders) | 1 (1) | 1 (1)
Aortic valve incompetence (Cardiac disorders) | 1 (1) | 2 (2)
Aortic valve stenosis (Cardiac disorders) | 8 (8) | 14 (14)
Arrhythmia (Cardiac disorders) | 0 (0) | 3 (5)
Arteriosclerosis coronary artery (Cardiac disorders) | 9 (9) | 8 (8)
Atrial fibrillation (Cardiac disorders) | 82 (84) | 76 (80)
Atrial flutter (Cardiac disorders) | 12 (13) | 13 (14)
Atrial tachycardia (Cardiac disorders) | 2 (2) | 4 (4)
Atrial thrombosis (Cardiac disorders) | 0 (0) | 1 (1)
Atrioventricular block (Cardiac disorders) | 2 (2) | 2 (2)
Atrioventricular block complete (Cardiac disorders) | 16 (16) | 18 (18)
Atrioventricular block first degree (Cardiac disorders) | 0 (0) | 1 (1)
Atrioventricular block second degree (Cardiac disorders) | 12 (12) | 6 (6)
Bifascicular block (Cardiac disorders) | 1 (1) | 0 (0)
Bradyarrhythmia (Cardiac disorders) | 2 (2) | 2 (2)
Bradycardia (Cardiac disorders) | 15 (15) | 6 (6)
Bundle branch block left (Cardiac disorders) | 1 (1) | 1 (1)
Bundle branch block right (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 7 (7) | 12 (12)
Cardiac disorder (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 64 (84) | 87 (108)
Cardiac failure acute (Cardiac disorders) | 20 (27) | 14 (15)
Cardiac failure chronic (Cardiac disorders) | 18 (19) | 30 (44)
Cardiac failure congestive (Cardiac disorders) | 60 (71) | 47 (53)
Cardiac tamponade (Cardiac disorders) | 0 (0) | 2 (2)
Cardiac valve disease (Cardiac disorders) | 0 (0) | 2 (2)
Cardiac ventricular scarring (Cardiac disorders) | 0 (0) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 3 (3) | 3 (3)
Cardiogenic shock (Cardiac disorders) | 6 (6) | 4 (4)
Cardiomyopathy (Cardiac disorders) | 1 (1) | 2 (2)
Cardiopulmonary failure (Cardiac disorders) | 1 (1) | 2 (2)
Cardiovascular insufficiency (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 85 (89) | 90 (95)
Coronary artery insufficiency (Cardiac disorders) | 2 (2) | 2 (2)
Coronary artery occlusion (Cardiac disorders) | 2 (2) | 2 (2)
Coronary artery stenosis (Cardiac disorders) | 14 (14) | 4 (4)
Dressler's syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Extrasystoles (Cardiac disorders) | 1 (1) | 0 (0)
Hypertensive heart disease (Cardiac disorders) | 0 (0) | 1 (1)
Ischaemic cardiomyopathy (Cardiac disorders) | 3 (3) | 2 (4)
Left ventricular dysfunction (Cardiac disorders) | 1 (1) | 1 (1)
Left ventricular failure (Cardiac disorders) | 7 (8) | 4 (4)
Microvascular coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1)
Mitral valve incompetence (Cardiac disorders) | 2 (2) | 3 (3)
Mitral valve stenosis (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial fibrosis (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 41 (43) | 65 (66)
Myocardial ischaemia (Cardiac disorders) | 36 (37) | 47 (50)
Myocarditis (Cardiac disorders) | 0 (0) | 1 (1)
Nodal arrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 4 (4) | 2 (2)
Pericardial effusion (Cardiac disorders) | 2 (2) | 1 (1)
Pericardial haemorrhage (Cardiac disorders) | 0 (0) | 1 (1)
Pericarditis (Cardiac disorders) | 3 (3) | 0 (0)
Pericarditis constrictive (Cardiac disorders) | 1 (1) | 1 (1)
Prinzmetal angina (Cardiac disorders) | 0 (0) | 3 (4)
Pulmonary valve incompetence (Cardiac disorders) | 0 (0) | 1 (1)
Right ventricular failure (Cardiac disorders) | 1 (1) | 2 (2)
Sinoatrial block (Cardiac disorders) | 0 (0) | 1 (1)
Sinus arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 7 (7) | 4 (4)
Sinus node dysfunction (Cardiac disorders) | 5 (5) | 4 (4)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 1 (1)
Stress cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1)
Supraventricular extrasystoles (Cardiac disorders) | 3 (3) | 2 (2)
Supraventricular tachycardia (Cardiac disorders) | 5 (5) | 9 (11)
Tachycardia (Cardiac disorders) | 1 (2) | 4 (4)
Tricuspid valve incompetence (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular arrhythmia (Cardiac disorders) | 1 (1) | 2 (2)
Ventricular asystole (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 4 (4) | 7 (7)
Ventricular fibrillation (Cardiac disorders) | 2 (2) | 3 (3)
Ventricular tachycardia (Cardiac disorders) | 10 (10) | 6 (6)
Corneal dystrophy (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Glucose-6-phosphate dehydrogenase deficiency (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Neurofibromatosis (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Deafness (Ear and labyrinth disorders) | 1 (1) | 2 (2)
Deafness neurosensory (Ear and labyrinth disorders) | 0 (0) | 2 (2)
Deafness unilateral (Ear and labyrinth disorders) | 3 (3) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Eustachian tube dysfunction (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Hypoacusis (Ear and labyrinth disorders) | 1 (1) | 1 (1)
Inner ear disorder (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Meniere's disease (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Sudden hearing loss (Ear and labyrinth disorders) | 2 (2) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Tympanic membrane perforation (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Tympanosclerosis (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 13 (13) | 7 (7)
Vertigo positional (Ear and labyrinth disorders) | 7 (7) | 3 (3)
Vestibular disorder (Ear and labyrinth disorders) | 2 (2) | 2 (2)
Adrenal insufficiency (Endocrine disorders) | 1 (1) | 0 (0)
Goitre (Endocrine disorders) | 5 (6) | 2 (2)
Hyperparathyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Hyperparathyroidism primary (Endocrine disorders) | 0 (0) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 2 (2)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Thyroiditis subacute (Endocrine disorders) | 1 (1) | 0 (0)
Age-related macular degeneration (Eye disorders) | 0 (0) | 1 (1)
Aphakia (Eye disorders) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 22 (26) | 30 (35)
Cataract cortical (Eye disorders) | 0 (0) | 1 (1)
Cataract diabetic (Eye disorders) | 0 (0) | 1 (1)
Cataract nuclear (Eye disorders) | 1 (1) | 1 (1)
Corneal degeneration (Eye disorders) | 1 (1) | 0 (0)
Diabetic retinopathy (Eye disorders) | 3 (5) | 4 (4)
Entropion (Eye disorders) | 0 (0) | 1 (1)
Eye haemorrhage (Eye disorders) | 4 (4) | 1 (1)
Eyelid ptosis (Eye disorders) | 1 (1) | 0 (0)
Glaucoma (Eye disorders) | 2 (2) | 3 (4)
Lacrimal disorder (Eye disorders) | 0 (0) | 1 (1)
Macular degeneration (Eye disorders) | 1 (1) | 1 (1)
Macular fibrosis (Eye disorders) | 2 (2) | 2 (2)
Macular oedema (Eye disorders) | 0 (0) | 1 (1)
Macular pseudohole (Eye disorders) | 1 (1) | 0 (0)
Maculopathy (Eye disorders) | 0 (0) | 1 (1)
Open angle glaucoma (Eye disorders) | 1 (1) | 0 (0)
Optic ischaemic neuropathy (Eye disorders) | 1 (1) | 0 (0)
Retinal artery occlusion (Eye disorders) | 1 (1) | 0 (0)
Retinal artery thrombosis (Eye disorders) | 0 (0) | 1 (1)
Retinal degeneration (Eye disorders) | 0 (0) | 1 (1)
Retinal detachment (Eye disorders) | 2 (2) | 3 (3)
Retinal haemorrhage (Eye disorders) | 2 (2) | 5 (5)
Retinal vein occlusion (Eye disorders) | 0 (0) | 1 (1)
Retinal vein thrombosis (Eye disorders) | 1 (1) | 0 (0)
Retinopathy (Eye disorders) | 0 (0) | 1 (1)
Retinopathy proliferative (Eye disorders) | 0 (0) | 1 (1)
Rhegmatogenous retinal detachment (Eye disorders) | 1 (1) | 0 (0)
Strabismus (Eye disorders) | 0 (0) | 1 (1)
Trichiasis (Eye disorders) | 0 (0) | 1 (1)
Ulcerative keratitis (Eye disorders) | 1 (1) | 0 (0)
Visual impairment (Eye disorders) | 1 (1) | 1 (1)
Vitreous haemorrhage (Eye disorders) | 9 (9) | 5 (5)
Vitreous opacities (Eye disorders) | 0 (0) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 2 (4) | 0 (0)
Abdominal hernia (Gastrointestinal disorders) | 2 (2) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 7 (7) | 4 (4)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 5 (5)
Abdominal wall haematoma (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anal fissure (Gastrointestinal disorders) | 0 (0) | 3 (3)
Anal fistula (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anal inflammation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Appendicitis noninfective (Gastrointestinal disorders) | 1 (1) | 0 (0)
Appendix disorder (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1)
Barrett's oesophagus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Bezoar (Gastrointestinal disorders) | 0 (0) | 1 (1)
Change of bowel habit (Gastrointestinal disorders) | 0 (0) | 1 (1)
Chronic gastritis (Gastrointestinal disorders) | 2 (2) | 4 (4)
Chronic gastrointestinal bleeding (Gastrointestinal disorders) | 1 (1) | 0 (0)
Coeliac disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 4 (4) | 5 (5)
Colitis ischaemic (Gastrointestinal disorders) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 4 (4) | 3 (3)
Dental caries (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diabetic gastroparesis (Gastrointestinal disorders) | 0 (0) | 1 (2)
Diaphragmatic hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 18 (18) | 8 (8)
Diverticular perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diverticulitis oesophageal (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diverticulum (Gastrointestinal disorders) | 3 (3) | 2 (2)
Diverticulum intestinal (Gastrointestinal disorders) | 4 (4) | 4 (4)
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 5 (6) | 2 (2)
Duodenal polyp (Gastrointestinal disorders) | 0 (0) | 1 (1)
Duodenal ulcer (Gastrointestinal disorders) | 4 (4) | 3 (3)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 7 (8) | 4 (4)
Duodenitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 3 (3) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 2 (2) | 3 (3)
Enteritis (Gastrointestinal disorders) | 2 (2) | 4 (4)
Enterocolitis (Gastrointestinal disorders) | 1 (1) | 2 (2)
Epigastric discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1)
Erosive oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Faecaloma (Gastrointestinal disorders) | 1 (1) | 1 (1)
Faeces discoloured (Gastrointestinal disorders) | 2 (2) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 2 (2)
Functional gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric antral vascular ectasia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric haemorrhage (Gastrointestinal disorders) | 6 (6) | 0 (0)
Gastric polyps (Gastrointestinal disorders) | 5 (5) | 6 (8)
Gastric ulcer (Gastrointestinal disorders) | 18 (18) | 9 (9)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 6 (6) | 3 (3)
Gastric ulcer perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 8 (8) | 12 (12)
Gastritis erosive (Gastrointestinal disorders) | 9 (9) | 2 (2)
Gastritis haemorrhagic (Gastrointestinal disorders) | 6 (6) | 1 (1)
Gastroduodenal ulcer (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastrointestinal angiodysplasia (Gastrointestinal disorders) | 2 (2) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 2 (2) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 43 (44) | 22 (23)
Gastrointestinal inflammation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal ischaemia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal motility disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal polyp haemorrhage (Gastrointestinal disorders) | 2 (2) | 1 (1)
Gastrointestinal stenosis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal ulcer haemorrhage (Gastrointestinal disorders) | 3 (3) | 2 (2)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 5 (6) | 7 (7)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 4 (4) | 2 (2)
Haemorrhagic erosive gastritis (Gastrointestinal disorders) | 1 (1) | 2 (2)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 3 (3) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 5 (5) | 2 (2)
Hernial eventration (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hiatus hernia (Gastrointestinal disorders) | 1 (1) | 2 (2)
Ileus (Gastrointestinal disorders) | 4 (5) | 3 (3)
Ileus paralytic (Gastrointestinal disorders) | 2 (2) | 0 (0)
Incarcerated inguinal hernia (Gastrointestinal disorders) | 1 (1) | 2 (2)
Inguinal hernia (Gastrointestinal disorders) | 16 (16) | 20 (20)
Intestinal haemorrhage (Gastrointestinal disorders) | 6 (6) | 3 (3)
Intestinal ischaemia (Gastrointestinal disorders) | 0 (0) | 3 (3)
Intestinal obstruction (Gastrointestinal disorders) | 4 (6) | 5 (5)
Intestinal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal polyp (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal pseudo-obstruction (Gastrointestinal disorders) | 1 (2) | 0 (0)
Intestinal strangulation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Large intestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Large intestine perforation (Gastrointestinal disorders) | 1 (1) | 2 (2)
Large intestine polyp (Gastrointestinal disorders) | 18 (18) | 14 (14)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 3 (3) | 3 (3)
Lumbar hernia (Gastrointestinal disorders) | 0 (0) | 2 (2)
Mallory-weiss syndrome (Gastrointestinal disorders) | 2 (2) | 1 (1)
Mechanical ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Melaena (Gastrointestinal disorders) | 12 (12) | 4 (4)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Obstruction gastric (Gastrointestinal disorders) | 1 (1) | 0 (0)
Obstructive pancreatitis (Gastrointestinal disorders) | 2 (2) | 2 (2)
Oesophageal motility disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophageal spasm (Gastrointestinal disorders) | 1 (2) | 0 (0)
Oesophageal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophageal ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 2 (2) | 1 (1)
Oesophagitis ulcerative (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatic mass (Gastrointestinal disorders) | 1 (1) | 1 (1)
Pancreatic pseudocyst (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 11 (14) | 7 (7)
Pancreatitis acute (Gastrointestinal disorders) | 2 (2) | 5 (6)
Pancreatitis chronic (Gastrointestinal disorders) | 4 (4) | 2 (2)
Pancreatolithiasis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Peptic ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Peptic ulcer haemorrhage (Gastrointestinal disorders) | 2 (2) | 0 (0)
Periodontal disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Peritoneal adhesions (Gastrointestinal disorders) | 0 (0) | 1 (1)
Peritoneal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Proctitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 13 (13) | 2 (2)
Rectal polyp (Gastrointestinal disorders) | 1 (1) | 1 (1)
Rectal prolapse (Gastrointestinal disorders) | 0 (0) | 1 (1)
Reflux gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Salivary gland calculus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal haemorrhage (Gastrointestinal disorders) | 2 (2) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 3 (3) | 4 (4)
Subileus (Gastrointestinal disorders) | 2 (2) | 1 (1)
Swollen tongue (Gastrointestinal disorders) | 0 (0) | 1 (2)
Tooth disorder (Gastrointestinal disorders) | 1 (1) | 1 (1)
Tooth socket haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ulcerative gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Umbilical hernia (Gastrointestinal disorders) | 4 (4) | 2 (2)
Umbilical hernia, obstructive (Gastrointestinal disorders) | 1 (1) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 22 (23) | 10 (10)
Varices oesophageal (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2) | 2 (2)
Administration site phlebitis (General disorders) | 1 (1) | 0 (0)
Asthenia (General disorders) | 4 (4) | 1 (1)
Capsular contracture associated with breast implant (General disorders) | 0 (0) | 1 (1)
Cardiac death (General disorders) | 4 (4) | 1 (1)
Catheter site haemorrhage (General disorders) | 1 (1) | 0 (0)
Chest discomfort (General disorders) | 5 (5) | 0 (0)
Chest pain (General disorders) | 6 (6) | 11 (11)
Complication associated with device (General disorders) | 0 (0) | 1 (1)
Death (General disorders) | 52 (52) | 60 (60)
Drowning (General disorders) | 1 (1) | 0 (0)
Facial pain (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 1 (1)
Foreign body reaction (General disorders) | 2 (2) | 0 (0)
Gait disturbance (General disorders) | 1 (1) | 1 (1)
Gait inability (General disorders) | 1 (1) | 0 (0)
General physical health deterioration (General disorders) | 2 (2) | 1 (1)
Impaired healing (General disorders) | 1 (1) | 1 (1)
Medical device site haemorrhage (General disorders) | 1 (1) | 0 (0)
Mucosal exfoliation (General disorders) | 1 (1) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 2 (2) | 0 (0)
Necrobiosis (General disorders) | 0 (0) | 1 (1)
Necrosis (General disorders) | 2 (2) | 2 (2)
Nodule (General disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 54 (60) | 66 (72)
Oedema (General disorders) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 1 (1) | 4 (4)
Pacemaker generated arrhythmia (General disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 8 (8) | 6 (6)
Sudden cardiac death (General disorders) | 6 (6) | 8 (8)
Sudden death (General disorders) | 5 (5) | 5 (5)
Ulcer haemorrhage (General disorders) | 1 (1) | 0 (0)
Vascular stent occlusion (General disorders) | 0 (0) | 1 (1)
Vascular stent stenosis (General disorders) | 6 (6) | 4 (5)
Acute hepatic failure (Hepatobiliary disorders) | 3 (3) | 0 (0)
Bile duct obstruction (Hepatobiliary disorders) | 2 (2) | 2 (2)
Bile duct stone (Hepatobiliary disorders) | 7 (7) | 3 (3)
Biliary colic (Hepatobiliary disorders) | 0 (0) | 1 (2)
Biliary dyskinesia (Hepatobiliary disorders) | 2 (2) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 1 (1) | 4 (5)
Cholangitis acute (Hepatobiliary disorders) | 3 (3) | 3 (3)
Cholangitis chronic (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 13 (14) | 23 (27)
Cholecystitis acute (Hepatobiliary disorders) | 19 (19) | 14 (15)
Cholecystitis chronic (Hepatobiliary disorders) | 5 (5) | 6 (6)
Cholelithiasis (Hepatobiliary disorders) | 23 (24) | 25 (25)
Cholestasis (Hepatobiliary disorders) | 0 (0) | 2 (2)
Chronic hepatitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cirrhosis alcoholic (Hepatobiliary disorders) | 0 (0) | 1 (1)
Drug-induced liver injury (Hepatobiliary disorders) | 0 (0) | 1 (1)
Gallbladder disorder (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic cirrhosis (Hepatobiliary disorders) | 4 (4) | 7 (7)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1) | 2 (2)
Hepatitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1)
Jaundice (Hepatobiliary disorders) | 0 (0) | 1 (1)
Jaundice cholestatic (Hepatobiliary disorders) | 1 (1) | 0 (0)
Liver injury (Hepatobiliary disorders) | 0 (0) | 1 (1)
Non-alcoholic steatohepatitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Portal vein thrombosis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Steatohepatitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Allergy to arthropod bite (Immune system disorders) | 1 (1) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 4 (4)
Anaphylactic shock (Immune system disorders) | 2 (2) | 1 (1)
Contrast media allergy (Immune system disorders) | 1 (1) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 4 (4)
Haemophagocytic lymphohistiocytosis (Immune system disorders) | 0 (0) | 1 (1)
Sarcoidosis (Immune system disorders) | 1 (1) | 0 (0)
Transplant rejection (Immune system disorders) | 0 (0) | 1 (1)
Abdominal abscess (Infections and infestations) | 1 (1) | 2 (2)
Abdominal sepsis (Infections and infestations) | 1 (1) | 0 (0)
Abdominal wall abscess (Infections and infestations) | 0 (0) | 1 (1)
Abscess jaw (Infections and infestations) | 1 (1) | 1 (1)
Abscess limb (Infections and infestations) | 5 (5) | 1 (1)
Abscess neck (Infections and infestations) | 0 (0) | 1 (1)
Acinetobacter infection (Infections and infestations) | 0 (0) | 1 (1)
Acute endocarditis (Infections and infestations) | 0 (0) | 1 (1)
Acute hepatitis b (Infections and infestations) | 0 (0) | 1 (1)
Acute sinusitis (Infections and infestations) | 1 (1) | 1 (1)
Anal abscess (Infections and infestations) | 3 (3) | 2 (2)
Anal fistula infection (Infections and infestations) | 0 (0) | 1 (1)
Appendiceal abscess (Infections and infestations) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 13 (14) | 10 (10)
Appendicitis perforated (Infections and infestations) | 3 (3) | 0 (0)
Arthritis infective (Infections and infestations) | 1 (1) | 0 (0)
Atypical pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 2 (2) | 1 (1)
Bacterial diarrhoea (Infections and infestations) | 0 (0) | 1 (1)
Bacterial sepsis (Infections and infestations) | 1 (1) | 0 (0)
Biliary sepsis (Infections and infestations) | 0 (0) | 1 (1)
Brain abscess (Infections and infestations) | 1 (1) | 0 (0)
Breast abscess (Infections and infestations) | 1 (1) | 0 (0)
Breast cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Bronchiolitis (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 18 (18) | 22 (23)
Bronchitis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Bursitis infective (Infections and infestations) | 1 (1) | 0 (0)
Campylobacter gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 35 (40) | 45 (51)
Cellulitis gangrenous (Infections and infestations) | 0 (0) | 2 (2)
Cellulitis of male external genital organ (Infections and infestations) | 1 (1) | 0 (0)
Cholangitis infective (Infections and infestations) | 2 (2) | 1 (1)
Cholecystitis infective (Infections and infestations) | 3 (3) | 2 (2)
Chronic hepatitis c (Infections and infestations) | 1 (1) | 2 (2)
Chronic sinusitis (Infections and infestations) | 1 (1) | 2 (2)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 1 (1)
Clostridium difficile infection (Infections and infestations) | 2 (2) | 3 (5)
Complicated appendicitis (Infections and infestations) | 1 (1) | 1 (1)
Cystitis (Infections and infestations) | 4 (4) | 4 (4)
Dacryocystitis (Infections and infestations) | 0 (0) | 1 (1)
Dengue fever (Infections and infestations) | 1 (1) | 1 (1)
Dengue haemorrhagic fever (Infections and infestations) | 0 (0) | 1 (1)
Device related infection (Infections and infestations) | 1 (1) | 1 (1)
Device related sepsis (Infections and infestations) | 2 (2) | 0 (0)
Diabetic foot infection (Infections and infestations) | 3 (4) | 3 (4)
Diabetic gangrene (Infections and infestations) | 1 (1) | 1 (1)
Diarrhoea infectious (Infections and infestations) | 2 (2) | 0 (0)
Diverticulitis (Infections and infestations) | 11 (12) | 4 (4)
Diverticulitis intestinal haemorrhagic (Infections and infestations) | 3 (3) | 2 (2)
Dysentery (Infections and infestations) | 0 (0) | 1 (1)
Ear infection (Infections and infestations) | 1 (1) | 0 (0)
Emphysematous cystitis (Infections and infestations) | 1 (1) | 0 (0)
Endocarditis (Infections and infestations) | 0 (0) | 5 (5)
Endophthalmitis (Infections and infestations) | 0 (0) | 1 (2)
Enteritis infectious (Infections and infestations) | 0 (0) | 1 (1)
Enterobacter pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Enterocolitis infectious (Infections and infestations) | 1 (1) | 0 (0)
Epididymitis (Infections and infestations) | 4 (4) | 0 (0)
Epiglottitis (Infections and infestations) | 1 (1) | 2 (3)
Erysipelas (Infections and infestations) | 12 (12) | 10 (13)
Escherichia urinary tract infection (Infections and infestations) | 2 (2) | 2 (2)
Eye infection viral (Infections and infestations) | 1 (1) | 0 (0)
Febrile infection (Infections and infestations) | 1 (1) | 0 (0)
Fungal infection (Infections and infestations) | 0 (0) | 1 (1)
Gangrene (Infections and infestations) | 5 (5) | 12 (13)
Gastroenteritis (Infections and infestations) | 14 (15) | 18 (19)
Gastroenteritis bacterial (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis salmonella (Infections and infestations) | 0 (0) | 3 (3)
Gastroenteritis viral (Infections and infestations) | 3 (3) | 2 (2)
Gastrointestinal infection (Infections and infestations) | 1 (1) | 0 (0)
Genitourinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Graft infection (Infections and infestations) | 0 (0) | 1 (1)
Groin abscess (Infections and infestations) | 0 (0) | 2 (2)
H1n1 influenza (Infections and infestations) | 0 (0) | 1 (1)
Helicobacter gastritis (Infections and infestations) | 0 (0) | 1 (1)
Helicobacter infection (Infections and infestations) | 1 (1) | 0 (0)
Hepatitis a (Infections and infestations) | 1 (1) | 0 (0)
Hepatitis c (Infections and infestations) | 2 (2) | 0 (0)
Hepatitis e (Infections and infestations) | 1 (1) | 0 (0)
Herpes ophthalmic (Infections and infestations) | 0 (0) | 1 (1)
Herpes virus infection (Infections and infestations) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 5 (5) | 5 (5)
Incision site abscess (Infections and infestations) | 1 (1) | 0 (0)
Infected bite (Infections and infestations) | 1 (1) | 0 (0)
Infected cyst (Infections and infestations) | 0 (0) | 1 (1)
Infected dermal cyst (Infections and infestations) | 1 (1) | 0 (0)
Infected skin ulcer (Infections and infestations) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 1 (1)
Infectious colitis (Infections and infestations) | 0 (0) | 1 (1)
Infectious pleural effusion (Infections and infestations) | 1 (1) | 1 (1)
Infective exacerbation of bronchiectasis (Infections and infestations) | 0 (0) | 2 (3)
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 1 (2) | 1 (1)
Influenza (Infections and infestations) | 8 (8) | 10 (10)
Joint abscess (Infections and infestations) | 1 (1) | 0 (0)
Kidney infection (Infections and infestations) | 0 (0) | 1 (1)
Labyrinthitis (Infections and infestations) | 0 (0) | 1 (1)
Liver abscess (Infections and infestations) | 1 (1) | 2 (2)
Localised infection (Infections and infestations) | 7 (8) | 7 (8)
Lower respiratory tract infection (Infections and infestations) | 4 (4) | 5 (5)
Ludwig angina (Infections and infestations) | 1 (1) | 0 (0)
Lung abscess (Infections and infestations) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 10 (12) | 6 (7)
Meningitis (Infections and infestations) | 0 (0) | 1 (2)
Meningitis bacterial (Infections and infestations) | 0 (0) | 1 (1)
Meningococcal infection (Infections and infestations) | 0 (0) | 1 (1)
Necrotising fasciitis (Infections and infestations) | 1 (1) | 1 (1)
Neutropenic sepsis (Infections and infestations) | 1 (1) | 0 (0)
Oesophageal candidiasis (Infections and infestations) | 0 (0) | 1 (1)
Ophthalmic herpes zoster (Infections and infestations) | 1 (1) | 0 (0)
Orchitis (Infections and infestations) | 5 (5) | 1 (1)
Osteomyelitis (Infections and infestations) | 14 (16) | 7 (8)
Osteomyelitis acute (Infections and infestations) | 1 (1) | 0 (0)
Osteomyelitis chronic (Infections and infestations) | 3 (3) | 0 (0)
Otitis media (Infections and infestations) | 1 (1) | 1 (1)
Otitis media acute (Infections and infestations) | 2 (2) | 0 (0)
Otitis media chronic (Infections and infestations) | 2 (2) | 0 (0)
Pancreas infection (Infections and infestations) | 1 (1) | 0 (0)
Papilloma viral infection (Infections and infestations) | 0 (0) | 1 (1)
Parainfluenzae virus infection (Infections and infestations) | 1 (1) | 0 (0)
Parotitis (Infections and infestations) | 2 (2) | 1 (1)
Perineal abscess (Infections and infestations) | 0 (0) | 1 (1)
Periodontitis (Infections and infestations) | 1 (1) | 1 (1)
Periorbital cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Peritonitis (Infections and infestations) | 3 (3) | 2 (2)
Peritonitis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Peritonsillar abscess (Infections and infestations) | 2 (2) | 1 (1)
Pharyngeal abscess (Infections and infestations) | 0 (0) | 2 (2)
Pneumocystis jirovecii infection (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 130 (137) | 147 (153)
Pneumonia bacterial (Infections and infestations) | 3 (3) | 3 (3)
Pneumonia escherichia (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia influenzal (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia mycoplasmal (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia staphylococcal (Infections and infestations) | 1 (1) | 1 (1)
Pneumonia streptococcal (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia viral (Infections and infestations) | 2 (2) | 1 (1)
Post procedural infection (Infections and infestations) | 2 (2) | 3 (3)
Post procedural sepsis (Infections and infestations) | 0 (0) | 1 (1)
Postoperative abscess (Infections and infestations) | 1 (1) | 0 (0)
Postoperative wound infection (Infections and infestations) | 3 (3) | 7 (7)
Prostatic abscess (Infections and infestations) | 1 (1) | 0 (0)
Prostatitis escherichia coli (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 8 (8) | 4 (4)
Pyelonephritis acute (Infections and infestations) | 3 (3) | 12 (12)
Pyelonephritis chronic (Infections and infestations) | 0 (0) | 2 (2)
Rectal abscess (Infections and infestations) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 4 (4) | 5 (5)
Respiratory tract infection viral (Infections and infestations) | 2 (2) | 1 (1)
Salmonellosis (Infections and infestations) | 0 (0) | 1 (1)
Scrotal abscess (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 14 (15) | 20 (20)
Septic shock (Infections and infestations) | 7 (7) | 7 (7)
Sinusitis (Infections and infestations) | 1 (1) | 2 (2)
Skin infection (Infections and infestations) | 0 (0) | 1 (1)
Soft tissue infection (Infections and infestations) | 0 (0) | 2 (2)
Staphylococcal infection (Infections and infestations) | 1 (1) | 1 (1)
Staphylococcal sepsis (Infections and infestations) | 1 (1) | 1 (1)
Streptococcal infection (Infections and infestations) | 0 (0) | 1 (1)
Streptococcal sepsis (Infections and infestations) | 4 (4) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 2 (3) | 1 (1)
Tonsillitis (Infections and infestations) | 1 (1) | 1 (1)
Tooth abscess (Infections and infestations) | 2 (2) | 1 (1)
Tracheobronchitis (Infections and infestations) | 0 (0) | 1 (1)
Tracheobronchitis mycoplasmal (Infections and infestations) | 1 (1) | 0 (0)
Tuberculosis (Infections and infestations) | 2 (2) | 0 (0)
Tuberculosis of genitourinary system (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 3 (3) | 5 (5)
Ureteritis (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 33 (37) | 36 (50)
Urinary tract infection bacterial (Infections and infestations) | 0 (0) | 1 (1)
Urosepsis (Infections and infestations) | 12 (13) | 10 (11)
Vestibular neuronitis (Infections and infestations) | 1 (1) | 1 (1)
Viral infection (Infections and infestations) | 2 (2) | 6 (6)
Vulval abscess (Infections and infestations) | 2 (2) | 0 (0)
Vulval cellulitis (Infections and infestations) | 1 (1) | 0 (0)
West nile viral infection (Infections and infestations) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 5 (5) | 4 (5)
Abdominal injury (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Accident at home (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Acetabulum fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Adrenal gland injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Anaemia postoperative (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Anastomotic leak (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Anastomotic stenosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 8 (8) | 8 (8)
Arterial bypass thrombosis (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Avulsion fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Brain contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Burns third degree (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Carbon monoxide poisoning (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Carotid artery restenosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Cataract traumatic (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Clavicle fracture (Injury, poisoning and procedural complications) | 1 (1) | 3 (3)
Concussion (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 7 (7) | 7 (7)
Coronary artery restenosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Coronary vascular graft occlusion (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Coronary vascular graft stenosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Craniocerebral injury (Injury, poisoning and procedural complications) | 5 (5) | 1 (1)
Dislocation of sternum (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Epidural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Extradural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Extraskeletal ossification (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Facial bones fracture (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Failure to anastomose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 5 (5) | 1 (2)
Femoral neck fracture (Injury, poisoning and procedural complications) | 3 (3) | 4 (4)
Femur fracture (Injury, poisoning and procedural complications) | 8 (8) | 15 (15)
Fibula fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 2 (2) | 4 (4)
Foreign body (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Foreign body in gastrointestinal tract (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fractured sacrum (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 8 (8) | 3 (3)
Heat stroke (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Hip fracture (Injury, poisoning and procedural complications) | 8 (8) | 9 (9)
Humerus fracture (Injury, poisoning and procedural complications) | 12 (12) | 8 (8)
Hyphaema (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Incisional hernia (Injury, poisoning and procedural complications) | 1 (1) | 3 (3)
Intervertebral disc injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Joint injury (Injury, poisoning and procedural complications) | 3 (3) | 4 (4)
Ligament injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ligament rupture (Injury, poisoning and procedural complications) | 4 (4) | 2 (2)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 12 (13) | 7 (8)
Lower limb fracture (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Lumbosacral plexus injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Median nerve injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 9 (9) | 5 (5)
Multiple fractures (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Multiple injuries (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Muscle injury (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Muscle strain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Nail injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Nerve injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Nerve root injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Nerve root injury lumbar (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Patella fracture (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Pelvic fracture (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Periorbital haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Periprocedural myocardial infarction (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Post procedural complication (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Post procedural fever (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural haematoma (Injury, poisoning and procedural complications) | 4 (4) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 11 (11) | 5 (5)
Postoperative ileus (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Postoperative respiratory failure (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Postoperative thoracic procedure complication (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Procedural complication (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Procedural haemorrhage (Injury, poisoning and procedural complications) | 2 (2) | 3 (3)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Pubis fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pulmonary contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Radiation pneumonitis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Radius fracture (Injury, poisoning and procedural complications) | 6 (7) | 8 (8)
Rib fracture (Injury, poisoning and procedural complications) | 4 (4) | 10 (10)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Scapula fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Seroma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Shunt malfunction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Skeletal injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skin injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 2 (2) | 6 (6)
Skull fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Skull fractured base (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spinal column injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 7 (7)
Spinal cord injury cervical (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Sternal fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Stomal hernia (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 23 (23) | 6 (6)
Subdural haemorrhage (Injury, poisoning and procedural complications) | 8 (8) | 5 (5)
Tendon injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 2 (2) | 8 (8)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Tibia fracture (Injury, poisoning and procedural complications) | 3 (3) | 6 (6)
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Traumatic fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Traumatic haematoma (Injury, poisoning and procedural complications) | 7 (7) | 2 (2)
Traumatic haemorrhage (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Traumatic haemothorax (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 11 (11) | 7 (7)
Ulna fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 6 (6) | 0 (0)
Urinary retention postoperative (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vascular graft complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Vascular graft thrombosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wound haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wound necrosis (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Wrist fracture (Injury, poisoning and procedural complications) | 2 (2) | 3 (3)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Bile output decreased (Investigations) | 1 (1) | 0 (0)
Blood follicle stimulating hormone increased (Investigations) | 1 (1) | 0 (0)
Blood glucose fluctuation (Investigations) | 1 (1) | 0 (0)
Blood glucose increased (Investigations) | 5 (5) | 3 (3)
Blood lactic acid increased (Investigations) | 0 (0) | 1 (1)
Blood potassium increased (Investigations) | 0 (0) | 2 (3)
Blood pressure increased (Investigations) | 2 (2) | 0 (0)
Blood urine present (Investigations) | 1 (1) | 0 (0)
Cardiac stress test abnormal (Investigations) | 3 (3) | 4 (4)
Electrocardiogram qrs complex prolonged (Investigations) | 0 (0) | 1 (1)
Electrocardiogram st segment depression (Investigations) | 1 (2) | 0 (0)
Electrocardiogram abnormal (Investigations) | 1 (1) | 0 (0)
Glycosylated haemoglobin increased (Investigations) | 1 (1) | 0 (0)
Haemoglobin decreased (Investigations) | 2 (2) | 3 (3)
Heart rate irregular (Investigations) | 1 (1) | 0 (0)
Hepatic enzyme increased (Investigations) | 1 (1) | 1 (1)
Hepatitis b surface antigen positive (Investigations) | 0 (0) | 1 (1)
Occult blood positive (Investigations) | 1 (1) | 0 (0)
Oxygen saturation decreased (Investigations) | 0 (0) | 1 (1)
Prostatic specific antigen increased (Investigations) | 2 (2) | 0 (0)
Troponin increased (Investigations) | 1 (1) | 2 (2)
Weight decreased (Investigations) | 2 (2) | 1 (1)
White blood cell count decreased (Investigations) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 6 (7) | 5 (5)
Diabetes mellitus (Metabolism and nutrition disorders) | 24 (28) | 42 (46)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 50 (55) | 60 (78)
Diabetic complication (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 10 (11) | 11 (13)
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 9 (9) | 17 (17)
Euglycaemic diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Fluid overload (Metabolism and nutrition disorders) | 2 (2) | 1 (2)
Gout (Metabolism and nutrition disorders) | 5 (7) | 6 (6)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 20 (21) | 22 (24)
Hyperglycaemic hyperosmolar nonketotic syndrome (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 5 (5) | 4 (4)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 33 (39) | 25 (26)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 5 (5) | 2 (2)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypovolaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Lactic acidosis (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Obesity (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 12 (12) | 19 (19)
Vitamin d deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (5) | 6 (6)
Arthritis (Musculoskeletal and connective tissue disorders) | 4 (4) | 5 (5)
Arthritis reactive (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 10 (11) | 14 (15)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (4)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Chest wall mass (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Chondromalacia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Compartment syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Crystal arthropathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Diabetic amyotrophy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Facial asymmetry (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Fistula (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Foot deformity (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 4 (4) | 5 (5)
Gouty tophus (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Inguinal mass (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (2)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 16 (17) | 19 (20)
Intervertebral disc space narrowing (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Joint contracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Loose body in joint (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 13 (13) | 7 (7)
Meniscal degeneration (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 9 (9) | 15 (15)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 9 (9)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Myofascitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myopathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Neuropathic arthropathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 47 (51) | 55 (57)
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteopenia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteorrhagia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (4) | 3 (3)
Patellofemoral pain syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3)
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Pseudarthrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 6 (6) | 3 (3)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 5 (5) | 8 (8)
Sacroiliitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Scoliosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Seronegative arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Sjogren's syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Soft tissue disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 8 (8) | 4 (4)
Spinal ligament ossification (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 6 (6) | 11 (12)
Spinal pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 1 (1)
Spondylitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Tendon disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Tenosynovitis stenosans (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Abdominal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 3 (3)
Acute promyelocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 1 (1)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 14 (14) | 6 (6)
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Adrenal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Adrenal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Anal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
B-cell lymphoma stage i (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (6) | 9 (10)
Benign gastric neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Benign neoplasm of bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Benign neoplasm of thyroid gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Benign ovarian tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 (8) | 9 (9)
Bladder cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 4 (4)
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 4 (4)
Bladder transitional cell carcinoma stage ii (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bone cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 1 (1)
Brain neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Breast cancer female (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9 (9) | 4 (4)
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 3 (3)
Breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Carcinoid tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cerebellopontine angle tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cervix carcinoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cervix carcinoma stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (4) | 1 (1)
Cholesteatoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Chordoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 1 (1)
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 4 (4)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 12 (12) | 16 (16)
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2)
Colorectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 4 (4)
Cutaneous lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Endometrial cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Endometrial cancer stage i (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Endometrial cancer stage ii (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Fibroadenoma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Fibrosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Fibrous histiocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Gallbladder adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Gallbladder adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Gallbladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Gallbladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Gastric adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 (7) | 10 (10)
Gastric neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Gastrointestinal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Gastrointestinal lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Gastrointestinal melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Gastrointestinal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Gastrointestinal stromal tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Gastrointestinal tract adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 4 (4)
Hepatic cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Hepatobiliary neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9 (10) | 4 (4)
Invasive breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Large intestine benign neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0)
Laryngeal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Lentigo maligna (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lip and/or oral cavity cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (3)
Lip neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lipofibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 6 (6)
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 14 (14) | 20 (20)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 (7) | 4 (4)
Malignant neoplasm of renal pelvis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Malignant neoplasm of unknown primary site (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Malignant neoplasm papilla of vater (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (2)
Meningioma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Metastases to peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastases to pleura (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastatic gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2)
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Monoclonal gammopathy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Muscle neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Musculoskeletal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 3 (3)
Nasopharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 3 (3)
Neoplasm prostate (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Non-hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 1 (1)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 4 (4)
Oesophageal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Oral neoplasm benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Osteoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2)
Ovarian fibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Ovarian granulosa cell tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Ovarian neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 12 (13) | 12 (12)
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Pancreatic neuroendocrine tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Pancreatic sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Papillary cystadenoma lymphomatosum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Penis carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Phyllodes tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pituitary tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 3 (3)
Plasmacytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Pleomorphic liposarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pleural neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 31 (31) | 36 (36)
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 4 (4)
Prostate cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Prostate cancer stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Prostate cancer stage iii (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 3 (3)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9 (9) | 3 (3)
Rectal cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Rectal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Rectosigmoid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Rectosigmoid cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 7 (7)
Renal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 3 (3)
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 3 (3)
Retroperitoneal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Salivary gland adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Salivary gland neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 2 (2)
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Small cell lung cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Small intestine adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Small intestine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Soft tissue sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 2 (2)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Squamous cell carcinoma of the cervix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Squamous cell carcinoma of the oral cavity (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Squamous cell carcinoma of the tongue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Thyroid adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 5 (5)
Thyroid cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Tongue neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2)
Tonsil cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Transitional cell cancer of the renal pelvis and ureter (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (5) | 1 (1)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Vulval cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Ageusia (Nervous system disorders) | 0 (0) | 1 (1)
Altered state of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Amnesia (Nervous system disorders) | 2 (2) | 0 (0)
Ataxia (Nervous system disorders) | 2 (2) | 0 (0)
Balance disorder (Nervous system disorders) | 0 (0) | 1 (1)
Basal ganglia haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Basal ganglia infarction (Nervous system disorders) | 0 (0) | 3 (3)
Brain hypoxia (Nervous system disorders) | 1 (1) | 0 (0)
Brain injury (Nervous system disorders) | 1 (1) | 0 (0)
Brain stem haemorrhage (Nervous system disorders) | 3 (3) | 0 (0)
Brain stem infarction (Nervous system disorders) | 1 (1) | 3 (3)
Brain stem stroke (Nervous system disorders) | 1 (1) | 0 (0)
Carotid arteriosclerosis (Nervous system disorders) | 0 (0) | 1 (1)
Carotid artery disease (Nervous system disorders) | 0 (0) | 2 (2)
Carotid artery occlusion (Nervous system disorders) | 3 (3) | 1 (1)
Carotid artery stenosis (Nervous system disorders) | 18 (18) | 21 (22)
Carotid sinus syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Carpal tunnel syndrome (Nervous system disorders) | 3 (3) | 3 (3)
Cauda equina syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Cerebellar haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Cerebellar infarction (Nervous system disorders) | 1 (1) | 0 (0)
Cerebellar stroke (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral arteriosclerosis (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral atrophy (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral haematoma (Nervous system disorders) | 1 (1) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 6 (6) | 6 (6)
Cerebral infarction (Nervous system disorders) | 18 (19) | 27 (28)
Cerebral ischaemia (Nervous system disorders) | 7 (9) | 3 (3)
Cerebral small vessel ischaemic disease (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 3 (3) | 9 (9)
Cerebrovascular insufficiency (Nervous system disorders) | 1 (1) | 2 (2)
Cervical cord compression (Nervous system disorders) | 0 (0) | 1 (1)
Cervical radiculopathy (Nervous system disorders) | 1 (1) | 2 (2)
Cervicobrachial syndrome (Nervous system disorders) | 0 (0) | 2 (2)
Cluster headache (Nervous system disorders) | 1 (1) | 0 (0)
Cognitive disorder (Nervous system disorders) | 0 (0) | 1 (1)
Coma (Nervous system disorders) | 0 (0) | 2 (2)
Dementia (Nervous system disorders) | 2 (2) | 4 (4)
Dementia with lewy bodies (Nervous system disorders) | 1 (1) | 0 (0)
Diabetic coma (Nervous system disorders) | 1 (1) | 0 (0)
Diabetic neuropathy (Nervous system disorders) | 9 (10) | 13 (14)
Dizziness (Nervous system disorders) | 14 (15) | 12 (12)
Dysarthria (Nervous system disorders) | 1 (1) | 0 (0)
Embolic cerebral infarction (Nervous system disorders) | 1 (1) | 1 (1)
Embolic stroke (Nervous system disorders) | 2 (2) | 1 (1)
Encephalopathy (Nervous system disorders) | 0 (0) | 2 (2)
Epilepsy (Nervous system disorders) | 1 (2) | 5 (7)
Epileptic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Essential tremor (Nervous system disorders) | 1 (1) | 0 (0)
Facial paralysis (Nervous system disorders) | 1 (1) | 3 (3)
Focal dyscognitive seizures (Nervous system disorders) | 1 (1) | 0 (0)
Generalised tonic-clonic seizure (Nervous system disorders) | 1 (1) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 1 (1) | 4 (4)
Haemorrhagic stroke (Nervous system disorders) | 10 (10) | 9 (9)
Haemorrhagic transformation stroke (Nervous system disorders) | 0 (0) | 3 (3)
Headache (Nervous system disorders) | 1 (2) | 2 (2)
Hemianopia (Nervous system disorders) | 1 (1) | 0 (0)
Hemiparesis (Nervous system disorders) | 2 (2) | 0 (0)
Hepatic encephalopathy (Nervous system disorders) | 2 (2) | 0 (0)
Hydrocephalus (Nervous system disorders) | 0 (0) | 2 (2)
Hypertensive encephalopathy (Nervous system disorders) | 5 (5) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 2 (2) | 1 (1)
Hypoglycaemic coma (Nervous system disorders) | 1 (1) | 1 (2)
Hypoglycaemic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Hypoglycaemic seizure (Nervous system disorders) | 1 (1) | 0 (0)
Hypoglycaemic unconsciousness (Nervous system disorders) | 0 (0) | 1 (1)
Iiird nerve paralysis (Nervous system disorders) | 0 (0) | 3 (3)
Intracranial aneurysm (Nervous system disorders) | 0 (0) | 1 (1)
Intracranial pressure increased (Nervous system disorders) | 0 (0) | 1 (1)
Ischaemic cerebral infarction (Nervous system disorders) | 0 (0) | 3 (3)
Ischaemic stroke (Nervous system disorders) | 85 (88) | 119 (127)
Lacunar infarction (Nervous system disorders) | 9 (10) | 5 (5)
Lacunar stroke (Nervous system disorders) | 0 (0) | 1 (1)
Loss of consciousness (Nervous system disorders) | 4 (4) | 4 (4)
Lumbar radiculopathy (Nervous system disorders) | 1 (1) | 2 (2)
Lumbosacral radiculopathy (Nervous system disorders) | 0 (0) | 1 (1)
Metabolic encephalopathy (Nervous system disorders) | 1 (1) | 2 (2)
Microsleep (Nervous system disorders) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 1 (1) | 1 (1)
Miller fisher syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Myasthenia gravis (Nervous system disorders) | 1 (1) | 0 (0)
Myelopathy (Nervous system disorders) | 0 (0) | 1 (1)
Nerve compression (Nervous system disorders) | 1 (1) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 1 (1)
Normal pressure hydrocephalus (Nervous system disorders) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Paralysis (Nervous system disorders) | 1 (1) | 1 (1)
Parkinson's disease (Nervous system disorders) | 1 (1) | 7 (8)
Parkinsonism (Nervous system disorders) | 0 (0) | 3 (3)
Peripheral nerve lesion (Nervous system disorders) | 1 (1) | 1 (1)
Petit mal epilepsy (Nervous system disorders) | 0 (0) | 1 (1)
Polyneuropathy (Nervous system disorders) | 2 (2) | 0 (0)
Post-traumatic headache (Nervous system disorders) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 5 (5) | 4 (4)
Pseudoradicular syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Putamen haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Radicular pain (Nervous system disorders) | 1 (1) | 0 (0)
Radiculopathy (Nervous system disorders) | 1 (1) | 2 (2)
Sciatica (Nervous system disorders) | 4 (4) | 9 (9)
Sedation (Nervous system disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 2 (2) | 6 (7)
Spinal cord compression (Nervous system disorders) | 0 (0) | 1 (1)
Spinal epidural haematoma (Nervous system disorders) | 0 (0) | 1 (1)
Subarachnoid haemorrhage (Nervous system disorders) | 2 (2) | 3 (3)
Syncope (Nervous system disorders) | 26 (29) | 27 (28)
Tension headache (Nervous system disorders) | 2 (2) | 0 (0)
Thalamic infarction (Nervous system disorders) | 0 (0) | 1 (1)
Thalamus haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Thoracic outlet syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Toxic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Transient global amnesia (Nervous system disorders) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 39 (39) | 33 (34)
Tremor (Nervous system disorders) | 0 (0) | 1 (1)
Vith nerve disorder (Nervous system disorders) | 0 (0) | 1 (1)
Vith nerve paralysis (Nervous system disorders) | 0 (0) | 1 (1)
Vith nerve paresis (Nervous system disorders) | 0 (0) | 1 (1)
Vascular dementia (Nervous system disorders) | 0 (0) | 2 (2)
Vascular encephalopathy (Nervous system disorders) | 1 (1) | 2 (2)
Vertebral artery dissection (Nervous system disorders) | 1 (1) | 0 (0)
Vertebral artery stenosis (Nervous system disorders) | 1 (1) | 0 (0)
Vertebrobasilar insufficiency (Nervous system disorders) | 2 (2) | 1 (1)
Vertigo cns origin (Nervous system disorders) | 2 (2) | 1 (2)
Device dislocation (Product Issues) | 2 (2) | 0 (0)
Device failure (Product Issues) | 0 (0) | 1 (1)
Device loosening (Product Issues) | 1 (1) | 1 (1)
Device malfunction (Product Issues) | 1 (1) | 3 (3)
Device occlusion (Product Issues) | 1 (1) | 1 (1)
Adjustment disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Affective disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 3 (3)
Bipolar disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Borderline personality disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Completed suicide (Psychiatric disorders) | 1 (1) | 1 (1)
Confusional state (Psychiatric disorders) | 3 (3) | 1 (2)
Delirium (Psychiatric disorders) | 3 (3) | 3 (3)
Delirium tremens (Psychiatric disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 6 (7) | 4 (4)
Depression suicidal (Psychiatric disorders) | 1 (1) | 0 (0)
Disorientation (Psychiatric disorders) | 2 (2) | 0 (0)
Illness anxiety disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Major depression (Psychiatric disorders) | 1 (2) | 1 (2)
Mental disorder (Psychiatric disorders) | 0 (0) | 1 (2)
Mental status changes (Psychiatric disorders) | 1 (1) | 1 (1)
Neuropsychiatric symptoms (Psychiatric disorders) | 0 (0) | 1 (1)
Suicide attempt (Psychiatric disorders) | 1 (1) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 56 (59) | 39 (43)
Azotaemia (Renal and urinary disorders) | 1 (1) | 0 (0)
Bladder neck obstruction (Renal and urinary disorders) | 0 (0) | 2 (2)
Bladder neck sclerosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Bladder outlet obstruction (Renal and urinary disorders) | 0 (0) | 2 (2)
Bladder tamponade (Renal and urinary disorders) | 1 (1) | 0 (0)
Calculus bladder (Renal and urinary disorders) | 3 (3) | 7 (7)
Calculus urethral (Renal and urinary disorders) | 0 (0) | 1 (1)
Calculus urinary (Renal and urinary disorders) | 6 (7) | 3 (3)
Chronic kidney disease (Renal and urinary disorders) | 9 (10) | 15 (15)
Cystitis haemorrhagic (Renal and urinary disorders) | 2 (2) | 0 (0)
Diabetic nephropathy (Renal and urinary disorders) | 6 (6) | 3 (3)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0)
End stage renal disease (Renal and urinary disorders) | 4 (4) | 3 (3)
Glomerulonephritis (Renal and urinary disorders) | 1 (1) | 0 (0)
Glomerulosclerosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 32 (33) | 13 (13)
Haemorrhage urinary tract (Renal and urinary disorders) | 1 (1) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 4 (4) | 7 (7)
Hypertensive nephropathy (Renal and urinary disorders) | 1 (1) | 0 (0)
Micturition disorder (Renal and urinary disorders) | 1 (1) | 0 (0)
Nephritic syndrome (Renal and urinary disorders) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 16 (19) | 21 (24)
Nephropathy toxic (Renal and urinary disorders) | 0 (0) | 1 (1)
Nephrotic syndrome (Renal and urinary disorders) | 1 (1) | 4 (4)
Pelvi-ureteric obstruction (Renal and urinary disorders) | 1 (1) | 0 (0)
Perinephritis (Renal and urinary disorders) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal artery arteriosclerosis (Renal and urinary disorders) | 0 (0) | 1 (2)
Renal artery occlusion (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal artery stenosis (Renal and urinary disorders) | 1 (1) | 2 (2)
Renal colic (Renal and urinary disorders) | 0 (0) | 2 (2)
Renal cyst (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal disorder (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 16 (17) | 15 (15)
Renal haemorrhage (Renal and urinary disorders) | 1 (1) | 1 (1)
Renal hypertension (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal impairment (Renal and urinary disorders) | 10 (10) | 8 (8)
Renal injury (Renal and urinary disorders) | 1 (1) | 1 (1)
Renal mass (Renal and urinary disorders) | 2 (2) | 1 (1)
Stress urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0)
Tubulointerstitial nephritis (Renal and urinary disorders) | 1 (1) | 2 (2)
Ureteric stenosis (Renal and urinary disorders) | 1 (1) | 1 (1)
Ureterolithiasis (Renal and urinary disorders) | 18 (20) | 13 (14)
Urethral haemorrhage (Renal and urinary disorders) | 1 (1) | 0 (0)
Urethral stenosis (Renal and urinary disorders) | 5 (5) | 0 (0)
Urinary bladder polyp (Renal and urinary disorders) | 1 (1) | 1 (2)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 4 (4) | 7 (7)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1) | 2 (2)
Acquired hydrocele (Reproductive system and breast disorders) | 0 (0) | 2 (2)
Acquired phimosis (Reproductive system and breast disorders) | 1 (1) | 2 (2)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 26 (26) | 21 (21)
Breast mass (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Cervical dysplasia (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Cervix disorder (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Cystocele (Reproductive system and breast disorders) | 2 (2) | 1 (1)
Endometrial atrophy (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Endometrial hyperplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Genital haemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Gynaecomastia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Ovarian cyst (Reproductive system and breast disorders) | 2 (2) | 1 (1)
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 1 (2) | 0 (0)
Prostatic fibrosis (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Prostatic haemorrhage (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Prostatic obstruction (Reproductive system and breast disorders) | 0 (0) | 2 (2)
Prostatism (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 7 (7) | 5 (5)
Prostatomegaly (Reproductive system and breast disorders) | 3 (3) | 1 (1)
Uterine fibrosis (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Uterine haemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Uterine polyp (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Uterine prolapse (Reproductive system and breast disorders) | 1 (1) | 2 (2)
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Vaginal prolapse (Reproductive system and breast disorders) | 3 (3) | 0 (0)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 6 (8) | 7 (7)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 11 (12) | 7 (7)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 14 (18) | 7 (9)
Asthmatic crisis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bronchial disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Choking (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 27 (41) | 41 (57)
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (3)
Diaphragmatic paralysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 35 (36) | 29 (29)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 8 (8)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Epiglottic cyst (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 20 (20) | 11 (12)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (2)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Idiopathic interstitial pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 3 (6) | 3 (3)
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (2)
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Mediastinal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Paranasal cyst (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 5 (6)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 16 (16) | 19 (19)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 10 (10) | 5 (5)
Pulmonary sarcoidosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary toxicity (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory alkalosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 8 (9) | 8 (8)
Restrictive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0)
Actinic elastosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3)
Dermal cyst (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Diabetic foot (Skin and subcutaneous tissue disorders) | 29 (32) | 18 (25)
Diabetic ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Ecchymosis (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Henoch-schonlein purpura (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Intertrigo (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Ischaemic skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Lichen planus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Myxoid cyst (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Necrobiosis lipoidica diabeticorum (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Prurigo (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin mass (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin necrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 7 (7) | 12 (12)
Stevens-johnson syndrome (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1)
Accelerated hypertension (Vascular disorders) | 1 (1) | 2 (2)
Air embolism (Vascular disorders) | 1 (1) | 0 (0)
Angiopathy (Vascular disorders) | 1 (1) | 0 (0)
Aortic aneurysm (Vascular disorders) | 8 (8) | 9 (9)
Aortic arteriosclerosis (Vascular disorders) | 0 (0) | 1 (1)
Aortic dissection (Vascular disorders) | 1 (1) | 0 (0)
Aortic stenosis (Vascular disorders) | 5 (5) | 7 (8)
Arterial occlusive disease (Vascular disorders) | 0 (0) | 2 (2)
Arterial stenosis (Vascular disorders) | 0 (0) | 1 (1)
Arterial thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Arteriosclerosis (Vascular disorders) | 0 (0) | 1 (1)
Artery dissection (Vascular disorders) | 0 (0) | 1 (1)
Atherosclerotic plaque rupture (Vascular disorders) | 1 (1) | 0 (0)
Blood pressure inadequately controlled (Vascular disorders) | 1 (1) | 0 (0)
Circulatory collapse (Vascular disorders) | 1 (1) | 3 (3)
Deep vein thrombosis (Vascular disorders) | 6 (6) | 8 (8)
Diabetic vascular disorder (Vascular disorders) | 1 (1) | 3 (3)
Embolism arterial (Vascular disorders) | 1 (1) | 0 (0)
Embolism venous (Vascular disorders) | 1 (1) | 0 (0)
Extremity necrosis (Vascular disorders) | 5 (6) | 1 (1)
Hypertension (Vascular disorders) | 36 (40) | 45 (45)
Hypertensive crisis (Vascular disorders) | 15 (17) | 23 (25)
Hypertensive emergency (Vascular disorders) | 4 (4) | 2 (2)
Hypotension (Vascular disorders) | 9 (10) | 6 (7)
Hypovolaemic shock (Vascular disorders) | 1 (1) | 1 (1)
Iliac artery disease (Vascular disorders) | 0 (0) | 1 (1)
Iliac artery embolism (Vascular disorders) | 0 (0) | 1 (1)
Intermittent claudication (Vascular disorders) | 9 (9) | 7 (8)
Labile blood pressure (Vascular disorders) | 0 (0) | 1 (1)
Lymphocele (Vascular disorders) | 1 (1) | 0 (0)
Lymphoedema (Vascular disorders) | 1 (1) | 0 (0)
Malignant hypertension (Vascular disorders) | 2 (2) | 0 (0)
Necrosis ischaemic (Vascular disorders) | 0 (0) | 1 (1)
Neurogenic shock (Vascular disorders) | 0 (0) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 7 (7) | 2 (2)
Peripheral arterial occlusive disease (Vascular disorders) | 31 (38) | 48 (60)
Peripheral artery aneurysm (Vascular disorders) | 1 (1) | 1 (1)
Peripheral artery occlusion (Vascular disorders) | 2 (2) | 2 (3)
Peripheral artery stenosis (Vascular disorders) | 10 (10) | 4 (4)
Peripheral artery thrombosis (Vascular disorders) | 5 (6) | 6 (6)
Peripheral coldness (Vascular disorders) | 0 (0) | 1 (1)
Peripheral embolism (Vascular disorders) | 0 (0) | 2 (2)
Peripheral ischaemia (Vascular disorders) | 14 (17) | 18 (19)
Peripheral vascular disorder (Vascular disorders) | 3 (3) | 5 (6)
Peripheral venous disease (Vascular disorders) | 3 (3) | 3 (3)
Rheumatoid vasculitis (Vascular disorders) | 0 (0) | 1 (1)
Shock (Vascular disorders) | 0 (0) | 2 (2)
Shock haemorrhagic (Vascular disorders) | 2 (2) | 0 (0)
Subclavian artery stenosis (Vascular disorders) | 1 (1) | 1 (1)
Subgaleal haematoma (Vascular disorders) | 1 (1) | 0 (0)
Temporal arteritis (Vascular disorders) | 1 (1) | 1 (1)
Thrombophlebitis (Vascular disorders) | 0 (0) | 1 (1)
Thrombophlebitis superficial (Vascular disorders) | 0 (0) | 2 (2)
Thrombosis (Vascular disorders) | 1 (1) | 1 (1)
Varicose vein (Vascular disorders) | 0 (0) | 1 (1)
Vascular compression (Vascular disorders) | 0 (0) | 1 (1)
Vascular occlusion (Vascular disorders) | 1 (1) | 0 (0)
Venous thrombosis limb (Vascular disorders) | 0 (0) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ticagrelor 60 mg (N=9562) | Ticagrelor Placebo (N=9531)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1951 (2479) | 610 (687)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2017-02-07): https://cdn.clinicaltrials.gov/large-docs/95/NCT01991795/Prot_000.pdf
  • Statistical Analysis Plan (2018-09-17): https://cdn.clinicaltrials.gov/large-docs/95/NCT01991795/SAP_001.pdf